

# HEALTHY MOM, HEALTHY BABY PPCC COUNSELOR TRAINING GUIDE

# **PPCC Counselor Training Guide**

# **Table of Contents**

| Chap | oter I - Introduction | 2 |
|------|------------------------------------------------------------|----|
| A. | What is the PPCC program? | 3 |
| В. | How does it work? | 3 |
| C. | PPCC Call Schedule | 4 |
| D. | Protocol for Calling Participants | 5 |
| Chap | oter II Basics of Counseling | 6 |
| A. | Informed Consent, Recording Permission, and Initial Intake | 7 |
| В. | Determining Readiness | 7 |
| C. | Establishing Goals | 7 |
| D. | Creating an Action Plan | 9 |
| E. | Providing Consistent and Ongoing support | 10 |
| F. | Tips for PPCC Counselors | 11 |
| Chap | oter III – PPCC Protocol for Changing Smoking Behavior | 12 |
| Α. | The Program | 13 |
| В. | Introduction Script | 13 |
| C. | Topic 1 – Introduction to PPCC | 15 |
| D. | Topic 2 – Baby's Birth | 20 |
| E. | Topic 3 – Understanding the Process of Behavior Change | 23 |
| F. | Topic 4 – Managing Day-to-Day Stress | 26 |
| G. | Topic 5 – Partner Support | 34 |
| Н. | Topic 6 – Breaking Down Common Barriers | 37 |
| I. | Topic 7 – The Quit Plan | 41 |
| J. | Topic 8 – Relapse Prevention | 49 |
| K. | Topic 9 – Eating Well and Staying Healthy | 54 |
| L. | Topic 10 – Maintaining a Tobacco-Free Life | 59 |
| Ap | pendix A: My Personal Quit Plan | 63 |
| Ap | pendix B: My Plan to Stay Tobacco-Free | 74 |
| Ap | pendix C: Approaches to Quitting Smoking | 76 |
| Ap | pendix D: Handling Difficult Questions and Statements | 87 |
| Ap | pendix E: Distressed Participant Protocol | 90 |



## A. What is the PPCC program?

Phone-Based Postpartum Continuing Care (PPCC), a.k.a. Healthy Mom, Healthy Baby (HMHB), is a supportive program designed to help women who have recently had a baby quit using tobacco products and/or stay quit. It consists of 10 calls over the course of 6 months, which will help the participant to maintain and/or implement her unique smoking cessation plan.

PPCC is currently being pilot-tested to determine its feasibility, acceptability, and efficacy. This study project is being funded by the National Institutes of Health.

Participants in this study are recruited from the Maryland Women's Center, a public obstetrics clinic in Baltimore, Maryland, during their first prenatal appointment. At the time of enrollment (typically in the first trimester of pregnancy), all reported having smoked regularly in the past year, currently smoking, or quitting within the past 90 days. During pregnancy, the women received the existing standard of care treatment (5 A's) during pregnancy from their physicians. The American College of Obstetricians and Gynecologists (ACOG, 2010) recommends the use of the 5 A's behavioral counseling framework to help pregnant women quit: Ask about tobacco use, Advise to quit, Assess willingness to make a quit attempt, Assist in quit attempt, and Arrange follow-up. PPCC incorporates the 5 A's into Chestnut Global Partners' existing phone-based tobacco cessation protocol, and adapts it for the postpartum period.

Your role as a PPCC Counselor is to help guide and support the study participants through the challenges of this process. Some of the women will have quit smoking during pregnancy, some will have cut down, and some will not have modified their smoking behaviors at all. Regardless, the postpartum period is very different than pregnancy, and a large majority of women return to their pre-pregnancy smoking behaviors within six months after giving birth. Not everyone will succeed the first time they try to quit. Some will need to come back several times before finding what works for them, and you can play an important role in their journey.

#### B. How does it work?

PPCC is a proactive program where a personal PPCC Counselor provides scheduled support calls to the participant, and encourages participants to call the 24/7 hotline if they are experiencing any urges/cravings or have a lapse or relapse to smoking.

Each of the 10 calls will assess current tobacco use, introduce a topic, and provide information that is useful in the maintenance or development of a tobacco cessation plan. Some calls will end with a weekly assignment designed to help the participant practice with and prepare for the new behaviors they will need to establish to become tobacco-free.

It is important to note that each woman may be at a different stage in the quitting process, and each call must be uniquely tailored to where she is. For example, the theme listed as topic 8 may be more appropriate to discuss in call 4. This booklet

does not need to be followed linearly. All themes should be discussed at some point during the 10 calls, but the order of the topics discussed is not critical.

You can support your client by becoming familiar with the modules and following up with your client at the scheduled times to discuss her progress. A sample call schedule appears below.

# C. PPCC CALL SCHEDULE

| | Sample call dates: |
|---|---|
| Call 1 – 36 weeks of pregnancy | 09/01/2013 |
| Call 2 – Within one week following the birth of the child (09/15/2013 | 09/22/2013 |
| Call 3 – 2 weeks after call 2 | 10/06/2013 |
| Call 4 – 2 weeks after call 3 | 10/20/2013 |
| Call 5 – 2 weeks after call 4 | 11/03/2013 |
| Call 6 – 2 weeks after call 5 | 11/17/2013 |
| Call 7 – 2 weeks after call 6 | 12/01/2013 |
| Call 8 – 1 month after call 7 | 01/01/2014 |
| Call 9 – 1 month after call 8 | 02/01/2014 |
| Call 10 – 1 month after call 9 | 03/01/2014 |

<sup>\*\*</sup>PPCC Counselor will be informed of the birth of the child within 48 hours.

<sup>\*\*</sup>Calls must be completed within 1 week of scheduled call date.

# D. PROTOCOL FOR CALLING PARTICIPANTS

# Calls for Sessions 1 and 2:

For Session 1 and Session 2, make daily attempts to reach the participant for two weeks (14 days). In the first week, call during the participant's best days/times between 3–5 times total each day and on any days not listed as "best days" 1-2 times each day. In the second week, call during both participant's best days/times and days/times not listed 3–5 times each day. Leave only one voicemail per day, if permission has been obtained from initial informed consent. Log all call attempts in the Call Log. If you have not been able to reach the participant after 2 weeks of call attempts, inform the PI and Project Coordinator (PC), who will attempt to contact the participant via email.

# Calls for Sessions 3 through 10:

For Sessions 3 through 10, call the participant at the scheduled call time, 5 minutes later, 10 minutes later, 25 minutes later, and 1 hour later (or whenever convenient for the Counselor based on her schedule), such that the Counselor makes at least 5 call attempts on the scheduled day, with at least 4 being in the first half hour of the scheduled time. After the scheduled day, make 3-5 call attempts daily for the first week, and 2-3 call attempts daily for the second week. Leave only one voicemail per day, if permission has been obtained from initial informed consent. Log all call attempts in the Call Log. If you have not been able to reach the participant after 1 week, inform the PI and PC, who will attempt to contact the participant via email; however, continue to make call attempts during week 2 unless you hear otherwise from the PI or PC.

\*\*Note that if you are able to make contact within 5 minutes of the scheduled time, you should have enough time to proceed with the call as planned. If you make contact with the participant 10 or 25 minutes after the scheduled time, you may need to reschedule if proceeding with the call would interfere with the next planned call. If you make contact with the participant later in the day, you may choose to either proceed with the session at that time if convenient for both parties, or you can simply reschedule the Session for a date that is within one week of the initial scheduled call.



# A. INFORMED CONSENT, RECORDING PERMISSION, AND INITIAL INTAKE

The first time you call the participant, informed consent should be read, recording permission should be obtained, and an initial intake should be completed.

Before each PPCC call, be prepared:

- Review the folder of the participant including her name, telephone number, and the date of the scheduled call.
- Have your schedule available (in case you need to reschedule an appointment).
- Have all materials needed for the call available.
- Encourage participant to follow along in her Healthy Mom, Healthy Baby Guide.
- Refer to Documentation Booklet once call begins to document all necessary information.

#### B. DETERMINING READINESS

The first step in helping your client create a plan is to determine their readiness to take on a behavior modification program. If a client is not ready to take on a significant behavior change, it is unlikely that they will be successful in quitting tobacco. The **Contemplation Ladder** (Biener & Abrams, 1991), located on page 1 of the Documentation Booklet, will help you to determine your client's current stage of readiness to quit smoking.

# C. ESTABLISHING GOALS

Once you have determined your client's readiness to make a behavior change, it is time to help her establish meaningful goals. You already know that her ultimate goal is to stop using tobacco products, but she will need to achieve smaller goals first.

When helping your client set goals, be aware of her stage of readiness. If someone is not ready to make concrete changes, the goals you suggest for her should reflect that.

Use the S.M.A.R.T goal system for helping to set useful goals as outlined below:

S.M.A.R.T. GOALS

**SPECIFIC** 

**MEASURABLE** 

**ATTAINABLE** 

REALISTIC

TIMELY

- **S. SPECIFIC:** A specific goal has a much greater chance of being achieved than a general goal. Use the six 'W's" to help create a specific goal.
- Who? Who is involved in the goal? Do you need to speak to others about your goal?
- What? What do you want to accomplish?
- Where? Where will the goal be achieved? Do you need to arrange a specific location for your goal?
- When? What date and time will the goal take place?
- Why? What is the purpose of the goal? What are your reasons for wanting to achieve your goal?
- Which? Are there any barriers or constraints to accomplishing your goal?

# M. MEASURABLE: Establish criteria for measuring the goal.

- How will you know when the goal has been reached?
- How will you measure your success or failure?

# A. ATTAINABLE: How will I attain my goal?

What is your step-by-step plan for reaching your goal

## R. REALISTIC:

- Are you willing to work towards this goal?
- Is the goal realistic considering your current circumstances?

# T. Timely:

- When will the goal be accomplished?
- Are there any barriers to meeting your deadline?

# Two Examples of tobacco-cessation goals:

1. A goal set without S.M.A.R.T. goals may look like this: "My goal is to quit smoking."

2. A goal set with S.M.A.R.T. goals may look like this:

"My goal is to cut back from 10 cigarettes a day to 5 cigarettes a day.

My deadline is May 1 for this goal.

I will talk to my partner and ask him to support me in this since he is also a smoker.

I will smoke my 5 cigarettes only when I am outside – I will not smoke at home, near the baby, within 30 minutes of breastfeeding, or in my car.

I want to achieve this goal because I know smoking is bad for my health and my baby's health, and I want to live a long, healthy life and be around for my grandchildren.

The biggest challenge for me will be not smoking with my friends, so I will go for a walk instead of smoking with them.

I will cut back from 10 cigarettes to 5 cigarettes gradually by smoking one less each day until I reach the goal of just 5 cigarettes each day.

I will call the 24/7 hotline whenever I feel an urge/craving to smoke or have a lapse/relapse, and will report on my progress to my PPCC Counselor during our scheduled calls."

## D. CREATING AN ACTION PLAN

An Action Plan is the step-by-step plan that your client will follow as she works to achieve her goals.

Each time you meet with your client, you should assess her stage of readiness and help her to set appropriate goals for the time between calls. The S.M.A.R.T. goals you set together will be the basis of her action plan.

Here is a sample action plan for a client who has just completed call 2 of the program.

#### Action Plan

# For client X

For September 22 - October 6

- 1. **ASSIGNMENT:** (from Topic 2 of the Program): List the steps you will take to protect your baby from secondhand smoke and nicotine that can be transmitted through breastfeeding.
- 2. **S.M.A.R.T GOALS:** This week you agreed to cut back from 10 cigarettes a day to 9 cigarettes a day. You will eliminate the cigarette you usually smoke right before breastfeeding in the morning. Instead of smoking, you will chew gum and listen to music on the radio. If you successfully meet this goal, you will treat yourself to dinner with your partner at the end of the week.
- 3. **NEXT APPOINTMENT:** Sunday, October 6 at 10:00 a.m. via phone
- 4. ADDITIONAL NOTES: Please call any time if you have questions or concerns this week!

#### E. PROVIDING CONSISTENT AND ONGOING SUPPORT

Successfully quitting the use of tobacco products is a process that is unique for each individual. Numerous factors influence her ability to quit including the amount of tobacco she uses, how long she has used it, how many of her family members and friends use tobacco, as well as other circumstances such as stress, fear of weight gain, and social pressures.

Because of the numerous and complex factors involved, consistent and ongoing support from the PPCC Counselor to the client is crucial.

- Schedule appointments at the set intervals with your clients.
- Make sure to follow-up with a client if she misses a scheduled appointment time with you, utilizing the protocol for reaching clients.
- Your client will need support as she alters her life to support this new change.
   Commit to long-term, consistent engagements with your client to discuss any challenges she is facing.
- Contact your client on her quit date to offer encouragement and support.

# RECOGNIZE THAT PREGNANT CLIENTS MAY DIFFER FROM NON-PREGNANT CLIENTS

- Participants in this study are typically low-income and African-American.
- They may have increased levels of stress due to the pregnancy itself and be under increased pressure to quit smoking for the health of the child.
- Participants are likely to have already cut down on their smoking prior to our first contact.
- The pregnancy may have initiated their first serious attempt to quit smoking.
- The woman may be ambivalent about the pregnancy and quitting smoking.

#### ENGAGE THE PARTICIPANT OVER THE PHONE

- Get to know her personal situation discuss her past quit attempts, specifically what worked and what did not work.
- Be sensitive to each caller's unique circumstances.
- Use critical listening skills and remain aware of changes in her voice, tone, sighs, and pauses and respond accordingly. Telephone counseling is like working "blind" – you must rely on all of your senses.
- Ask open-ended questions to encourage her to explain her answers.
- Use reflection and the five principles of motivational style of counseling: express empathy, develop discrepancy, avoid argumentation, roll with resistance, and support self-efficacy.
- If you hear background noise or the woman appears to be busy, offer to call back at a more convenient time.

#### UNDERSTAND BARRIERS SPECIFIC TO PREGNANT WOMEN

- Recognize that most pregnant women feel extremely guilty about smoking. Allow the women to talk about their guilt and tell them that participating in this program is an important step in quitting and demonstrates their strength.
- Emphasize what the women can do to quit smoking and don't focus on the difficulties of quitting.
- Realize that counseling can be hard for women who live with smokers.
- The women's physical and mental health during the pregnancy may be a barrier to quitting –let the women talk about this.
- Discuss cravings and challenges she may experience while quitting and tell her that a slip is not a failure.
- She may have little to no support.
- If the woman has been pregnant before and had a healthy baby, she may not comprehend the need to quit.
- Listen for signs of depression, domestic violence, or other crisis. Refer her to appropriate community resources and/or urge her to talk to a healthcare provider.



## A. THE PROGRAM

The 10 calls of the Program are designed to help you guide the study participant through the process of quitting tobacco as well as encouraging continued abstinence if she quit during pregnancy. The first weeks should be used to design a unique plan for each individual and to allow her to practice some of the behaviors she will need to adopt in order to achieve a successful guit.

# B. INTRODUCTION SCRIPT

| "Hi, my name is | and I'm calling from Healthy Mom, Healthy Ba | aby |
|---|---|---|
| May I speak with [FIRST NAME]?" | | - |

IF PARTICIPANT IS NOT AVAILABLE: "When would be a good time to call again?"

IF PARTICIPANT IS AVAILABLE: "A few months ago, you agreed to take part in a study about smoking cessation from pregnancy through postpartum at the Maryland Women's Center. I have been assigned to be your Counselor. My name is \_\_\_\_\_ and I will be calling you every couple of weeks for the next few months to check in with you to see how things are going and how I might help you cut down or quit smoking. Is now a good time to start?"

IF YES, CONTINUE READING INFORMED CONSENT.
IF NOT A GOOD TIME, RESCHEDULE WITH PARTICIPANT.

#### **INFORMED CONSENT**

# (TO BE READ AT CALL 1 ONLY)

Before we begin, I would like to remind you of the study details. The National Institutes of Health is funding this study, and it is designed to improve the treatment and support pregnant smokers receive at the Maryland Women's Center. As part of the study, we are offering smoking cessation counseling to women who are about to give birth and have given birth recently, and determining how helpful it is offer phone counseling during this time.

One goal of this study is to help women who have just had babies learn more about how smoking is unhealthy for mothers and babies, deal with cravings to smoke, and encourage them to quit smoking if they have started smoking again after the baby is born. As your Counselor, I will call you ten times over a six-month period to discuss things known to be associated with smoking, such as mood and stress and partner support. I will also offer suggestions on how to reduce the risks of transmitting nicotine (the addictive drug in cigarettes) to your infant through breastfeeding while smoking or smoking in his/her presence. Each call is expected to take 15-30 minutes, and you are encouraged to call in at any time if you are having cravings or would like the support of your Counselor at this number: 1-855-611-HMHB (4642).

# "Do you have any questions about anything I've said so far?"

#### **RECORDING PERMISSION**

(TO BE READ IN ITS ENTIRETY BEFORE CALL 1;

# ONLY BOLDED TEXT NEEDS TO BE READ AT START OF SUBSEQUENT CALLS)

In order to ensure that I am conducting this call accurately and properly, I would like to make an electronic audio recording of this call. This is done strictly for quality control purposes. The recording will only be listened to by staff members on the project who have signed confidentiality pledges. The recording will be stored in a secure manner and will not contain your name—only a random number that will be assigned to this case. To help maintain confidentiality, we ask that you not give your last name or any other identifying information, such as an address or place of business, during the call. All recordings will be permanently destroyed within twelve months after the end of the data collection period. We can still continue the call if you do not want me to record it.

Do you agree to allow me to record the call?

YES: "I will now begin recording." START RECORDING AND SAY: "This is [YOUR FIRST NAME] conducting telephone call [# of current telephone call] with Participant [RESEARCH ID] on [DATE]."

NO: DON'T RECORD "Ok, let's get started."

PROCEED TO CALL

Coaches Notes: Your first meeting with your client is an important time to prepare her for what is to come and to build a relationship with her.

- Establish rapport, then inquire about smoking status and quit date to determine how best to tailor the call.
- Complete an Initial Intake (see Documentation Booklet, p. 2) with your client to learn more about her health and tobacco use history. The goal of the intake is to acquire information about the participant's past and current behaviors in order to better customize her tobacco-cessation plan.
- Briefly review the call themes/topics of the program with her.
- Review Topic 1 with your client and create an action plan.
- Make sure you leave plenty of time for your client to ask questions about how the program will work and to express any fears or concerns she may have about quitting or staying quit after her baby is born.
- Document all information obtained in the Documentation Booklet.

First, I want to congratulate you on your pregnancy and in taking a major step on your path to getting healthier for you and your baby! How much are you smoking now? [If still smoking: Have you set a guit date? I want you to know that I am here to help you guit smoking whenever you are ready.]

Additional sample questions you may ask to build rapport:

How has your pregnancy been so far? Do you know if you're having a boy or a girl? Do you have a name picked out?

You should have received a booklet entitled "Healthy Mom, Healthy Baby" to follow along and make notes from our calls. Did you receive that? Do you have it with you now? (Document in Documentation Booklet)

For this first call, you'll be introduced to the program and review the costs of continuing and benefits of quitting smoking.

You may have tried to guit in the past, and it's important to look at those attempts as learning lessons rather than failures. You can guit smoking by taking it one day at a time. This program will help answer questions like: What triggered me to start smoking again after I guit?: What can I do differently this time?; and How can I handle stressful situations in the future, without smoking? The program will also prepare you for the various situations when getting ready to quit, when you actually quit, and when faced with an urge to smoke again.

Women are more likely to guit smoking during pregnancy than at any other time of their lives because they want to have a healthy baby. However, smoking after giving birth is also associated with risks to the baby and many women begin smoking again after having their baby.

This 10-call program is designed to help you build the confidence to succeed after your baby is born, including a solid plan to quit smoking and/or stay quit.

Included in your Healthy Mom, Healthy Baby Guide is a brief summary of the topics we will be covering as part of the program. I won't go into them in detail since you have them, but briefly: (Coaches Note: read call theme/topic only)

- **Topic 1 Introduction to Healthy Mom, Healthy Baby:** For this first week, you'll be introduced to the 10-call program in preparation for developing your personal quit or stay-quit plan. You will also look at the costs and benefits associated with your tobacco use to help you think about the reasons why you want to quit or stay quit. **Topic 2 Baby's Birth:** This call will focus on the impact the birth of your baby can have on smoking behaviors. We will discuss the health implications of returning to smoking postpartum for both you and your newborn, and identify strategies to avoid
- **Topic 3 Understanding the Process of Behavior Change:** This call will help you have a better understanding of what is involved with the process of making this significant lifestyle change.

relapse during this wonderful but stressful time.

- **Topic 4 Managing Day-to-Day Stress:** Stress may be a contributing factor to why you use tobacco. This call will teach you tobacco-free stress management skills for dealing with stress at home, work, and with everyday life.
- **Topic 5 Partner Support:** A partner can be helpful in encouraging you to quit smoking or can be harmful if he/she smokes around you and brings on an urge for you to smoke. This call focuses on how to speak with your partner about smoking and develop a plan for how to get the support you need.
- **Topic 6 Breaking down Common Barriers:** We will review some of the everyday barriers and challenges that can arise when quitting tobacco as well as strategies to overcome them.
- **Topic 7 The Quit Plan:** PPCC focuses heavily on both preparation for quitting and helping you work through any challenges for staying quit. In this call, you will have the opportunity to develop your personal quit plan or solidify your existing plan.
- **Topic 8 Relapse Prevention:** This call will help you determine the difference between a lapse and a relapse, and discusses approaches for managing both. Common obstacles to staying quit are identified and tips to overcome them are given.
- **Topic 9 Eating Well and Staying Healthy:** Taking care of yourself is essential to helping you stay quit. This call will review basic nutrition and fitness guidelines including tips for minimizing post-tobacco use weight gain.
- **Topic 10 Maintaining a Tobacco-Free Lifestyle:** Achieving a tobacco-free life is a significant and positive change to your overall health. However, living your healthiest life requires a look at the whole picture. With this program coming to an end, call 10 helps you create a concrete plan for remaining tobacco-free, and includes tips so you can continue this positive journey on your own.

After this call and the next, if there is a particular issue or topic you'd like to cover during a call, please let me know at the beginning of the call and we can focus on that topic. It is important to go through all of the topics, but they don't need to be in order.

At the beginning of each call, I'll ask you about your current tobacco use, assist you with managing any problems that came up since we last spoke, and acknowledge success in meeting goals. At the end of each call, we'll work together to develop an action plan for small goals you can meet in the time between our calls. Achieving these small goals will empower you and help you feel more in control of your life.

Now I'd like to get to know you a bit better so I have a better sense of how to help you. It's important that you feel comfortable talking with me too, and I want to be sure to give you the opportunity to ask any questions that you may have. I want you to know that you can stop me at any time if something isn't clear, if you want me to repeat something, or if you want to make a comment.

# PROCEED TO INTAKE (DOCUMENTATION BOOKLET)

I would like to briefly review some of the costs and benefits of quitting smoking. These are also included in your Healthy Mom, Healthy Baby Guide. Please remember that I am here to support you, not judge you and want to review this information with you so you are aware of the costs and benefits of quitting smoking.

What have you heard about the health impact of smoking during pregnancy?

\*\*Document in Documentation Booklet\*\*

# **COSTS/BENEFITS**

# Why Quit?

Quitting smoking not only reduces risks of health problems for the baby and complications during delivery but also benefits a woman's long-term health. Smoking is associated with many health risks for women, including:

- Cardiovascular disease Most coronary heart disease among women younger than 50 is attributable to smoking.
- Lung cancer Lung cancer surpassed breast cancer as the leading cause of cancer death in women in 1987. About 90% of all lung cancer deaths among U.S. women smokers are attributable to smoking.
- Premature death The annual risk for death from all causes is about 80-90% greater among women who smoke compared with those who have never smoked. For every death attributable to smoking, an average of 14 years of life is lost.

# When you stop smoking...

- Your baby will get more oxygen, even after just one day of not smoking.
- Your baby is less likely to have bronchitis and asthma.
- There is less risk that your baby will be born too early.
- There is a better chance that your baby will come home from the hospital with you.
- You will be less likely to develop heart disease, stroke, lung cancer, chronic

lung disease, and other smoke-related diseases.

- You will be more likely to live to know your grandchildren.
- You will have more energy and breathe more easily.
- You will have more money that you can spend on other things.
- Your clothes, hair, and home will smell better.
- Your food will taste better.
- You will feel good about what you have done for yourself and your baby.

#### TIMING OF HEALTH BENEFITS AFTER QUITTING SMOKING

| 20 minutes | Your heart rate drops. |
|---|---|
| 12 hours | Carbon monoxide level in your blood drops to normal. |
| 2 weeks to 3 months | Your heart attack risk begins to drop. Your lung function begins to improve. |
| 1 to 9 months | Your coughing and shortness of breath decrease. |
| 1 year | Your added risk of coronary heart disease is half that of a smoker's. |
| 5 to 15 years | Your stroke risk is reduced to that of a nonsmoker's. |
| 10 years | Your lung cancer death rate is about half that of a smoker's. Your risk of cancers of the mouth, throat, esophagus, bladder, kidney, and pancreas decreases. |
| 15 years | Your risk of coronary heart disease is back to that of a nonsmoker's. |

These are just some of the costs of continuing and benefits of quitting smoking.

# Which costs/benefits are the most important for you?

Document in Documentation Booklet

Okay, these are really important for us to keep in mind moving forward, because we can always go back and look at these when you feel the urge to smoke.

# What do you see as the biggest barriers you will face to quitting/staying quit once your baby is born?

Document in Documentation Booklet

Those do make it challenging, but we will work together over the next few weeks to figure out ways to overcome those barriers.

I know that quitting smoking and staying quit takes a lot of effort, but it will ultimately be the healthiest choice for you and your baby.

**Action Plan:** I mentioned before that we will develop an action plan at the end of each call for you to work on until we talk again. For this time, please try to write down when you feel the urge to smoke and what works and doesn't work to get you through the craving. You might pick a certain time of day (e.g., right before bed) to do this if it's not convenient to make note of cravings in the moment.

The other part of the action plan is developing a goal. Here's an example: "I will cut back from 10 cigarettes a day to 5 cigarettes a day. I will not smoke the cigarette I usually smoke right when I wake up in the morning or when I drive. Instead of smoking, I will chew gum and listen to music on the radio. If I successfully meet this goal, I will treat myself to dinner with my partner." What is your personal goal?

Document in Documentation Booklet

Great! I will give you a call again within the week after your baby is born. (The Maryland Women's Center will let us know when that is.) Please remember that any time you have the urge to smoke or are craving a cigarette, you can call our 800-number 24 hours a day 7 days a week and someone will be available to talk with you about your cravings and try to help identify other things you can do instead of smoking.

Before we hang up, I just want to verify the phone number to call for our next session:

\*Document in Documentation Booklet\*

Is it okay to leave a message on your voicemail if you are not available?

\*Document in Documentation Booklet\*

Thank you. I'll be calling you again soon after your baby is born. Do you have any questions before we end our call? I look forward to speaking with you again soon.

#### D. TOPIC 2 - BABY'S BIRTH

Congratulations on the birth of your baby!

[To further rapport-building, ask participant questions such as: the baby's name, how delivery went and how she's feeling, if she's nursing, etc.]

On this call we'll talk about the impact of smoking on your new baby, as well as how to avoid returning to the level of smoking you had prior to getting pregnant.

#### **Documentation**

Go to the Documentation Booklet to complete initial questions.

#### THE IMPACT OF SMOKING ON NEWBORNS

Children exposed to secondhand smoke have higher rates of upper respiratory infections, colds, and asthma. They also have a higher risk of sudden infant death syndrome (SIDS). Because their bodies are developing, poisons in smoke hurt babies even more than adults. Babies under a year old are in the most danger.

# If you do smoke, what are some ways you can reduce your baby's exposure to secondhand smoke?

**Document in Documentation Booklet** 

(If not mentioned)

Other ways you can lessen your baby's exposure to secondhand smoke are:

- Don't smoke in the house with the baby.
- Don't allow others to smoke in the same room as the baby.
- If you do smoke in your home, designate one room to be the smoking room and do not allow baby access to that room.

# Are you breastfeeding?

Document in Documentation Booklet

(If Yes, encourage the client to continue breastfeeding. If No, state that you would still like to let her know the following...)

Doctors emphasize the importance of breastfeeding, and information is included in your Healthy Mom, Healthy Baby Guide about how breastfeeding protects babies and benefits you as a mother.

# Did you know?

A breastfeeding mother who smokes transmits nicotine (the addictive drug in cigarettes) to her infant through her breast milk in concentrations between 1.5 and 3 times what she is experiencing.

# What are some ways you can make sure your baby doesn't get nicotine through your breast milk?

Document in Documentation Booklet

# (If not mentioned)

Other ways you can minimize the transmission of nicotine to your baby through breast milk are:

- Resolve to quit smoking until you have stopped breastfeeding.
- If you do smoke, don't smoke 30 minutes prior to breastfeeding.

There are many benefits of breastfeeding, and it is best if you can continue to breastfeed until your baby is one year old.

Many women either cut down or quit smoking during pregnancy but start smoking again at the pre-pregnancy levels in the first few weeks after giving birth. I want to briefly go over some tips for how to avoid this trap.

# Tips to avoid starting smoking after baby is born: (For women who quit smoking or cut down during pregnancy)

- ✓ Review your reasons for quitting/cutting down
- ✓ Think about how smoking may negatively affect your baby's health
- ✓ Ask your Counselor for strategies to deal with triggers
- ✓ Call your Counselor for personal support or encouragement

# Tips to deal with a lapse:

- ✓ Don't wait to take action, a slip can easily lead to a relapse
- ✓ Stop using tobacco immediately and throw away all tobacco and related items
- ✓ Remove yourself from the situation that led you to smoke.
- ✓ Evaluate what led to the slip: Where were you? Who were you with? What were you doing? How were you feeling?

# Remember, you have not failed and you can overcome a slip!

Do you have any questions before we move on to your action plan for next time?

Action Plan: For this time, please track your tobacco use. You can use the Smoking Tracker form in the back of your Healthy Mom, Healthy Baby Guide and use separate sheets if you need additional paper. If you smoke, make a note of the time of day, how badly you needed to smoke, and what you were feeling at the time. Please also make a note of where you were in relation to the baby when you smoked, including if you were breastfeeding within 30 minutes of smoking.

I will give you a call again in about two weeks. Do you know which topic you'd like to discuss next time? What is your personal goal for the next two weeks?

Document in Documentation Booklet

Please remember that any time you have the urge to smoke or are craving a cigarette, you can call our toll-free number 24 hours a day 7 days a week and someone will be

available to talk with you about your cravings and try to help you to identify other things you might do instead of smoking.

What would be the best date and time to call for our next session?

Document in Documentation Booklet

Could you also verify the phone number to call?

Document in Documentation Booklet

Thank you. Do you have any questions for me before we end our call? I look forward to speaking with you again soon.

# Rapport-Building

Begin by asking the participant how she and the baby are doing.

#### **Documentation**

Go to the Documentation Booklet to complete initial questions. Based on responses, choose a topic theme to discuss from the list. If the participant is still smoking at all, continue with topic 3. If it is unclear which topic to proceed with, you may ask the participant which may be most helpful for her at this time.

Coaches Notes: There are similar steps that must be taken to make any significant behavior change, and this call will help your client understand why you will be asking her to do many of the activities in this program. By making appropriate changes in routines, habits and rituals, your client will be setting herself up for success. You can support her in this by encouraging her to actively participate in all assignments throughout the program and by reminding her that practicing new behaviors will help her when her quit day arrives.

# **Understanding the Process of Behavior Change**

Quitting smoking is not a simple process, and especially not when you're dealing with a new baby. It requires looking at your behaviors and understanding other things that must change in your life in order to quit smoking. This call will help you have a better understanding of what is involved in making this lifestyle change.

For most of us, making a behavior change begins with setting a goal. We know what we want to accomplish and that is an important first step. However, developing a plan, making sure you can reach your goal, and creating support systems are essential to your ultimate success. This call will help you focus on the steps you will need to take on your road to guitting smoking.

# **Desire to Change**

There may be many areas of your life where you feel you could make improvements and one of the first steps in actually doing so is deciding where you really want to focus your energy. No matter who you are, everyone is striving to change or improve their lives in one way or another. Whether it's to lose weight, make more money, get better at doing something, or stop smoking, the desire is there for each and every one of us.

Question: What changes do you want to make in your life? How confident are you that you can make these changes?

Document in Documentation Booklet

One of the changes that we're focused on is helping you to quit smoking and stay quit. So now we'll talk about factors that influence your smoking.

# **Recognize Factors associated with Smoking**

The focus of this program is to identify the unhealthy behavior of smoking and replace this behavior, and any associated unhealthy behaviors, with healthy behaviors that will make you feel good and provide you with a way to be successful long-term.

Question: What are some things that you associate with your smoking?

#### **Self-Awareness**

You are on the path to quitting smoking and it's important to become aware of the people, places, and situations that play a role in your smoking. Smoking is associated with various everyday tasks. Becoming aware of why you smoke and how you are using tobacco to cope with certain problems is an important part of your success.

Question: Why do you smoke and how are you using smoking to deal with problems in your life?

# **Establishing Your Support**

Participation in this 10-call program is just one form of support for you through the quit process. The more support you can have, the more successful you'll be. Informing your co-workers, friends, and family that you're planning to quit smoking will provide you with accountability and plenty of people to turn to when the road gets difficult. Do you have friends or relatives from whom you can get support? [If yes, encourage participant to turn to them for support when they need it. If no, tell them: "You are not alone in this process and not the only one out there who has decided to quit. There are counselors, support groups and online resources available to help you through the process too."

Question: Have you had to approach others to help you get through something in the past? Who did you ask? How did this help?

# **Developing a Plan and Establishing Realistic Goals**

The idea of this step-by-step process is to approach your goal of quitting smoking with a well thought out plan and realistic goals to get you there. Short-term goals such as one less smoke break each day or not smoking in the car, will lead you to your long-term goal of being tobacco-free. This is what we've been doing with our Action Plan. Once you reach one goal, you can move towards your next and this will keep you feeling encouraged by your achievements along the way.

**Action Plan:** Create a list of people you feel comfortable talking to about your journey to quit smoking and who you feel would be encouraging, and call one when you feel like you need support or have the urge to smoke.

Also remember that any time you have the urge to smoke or are craving a cigarette, you can call our toll-free number 24 hours a day 7 days a week and someone will be available to talk with you about your cravings and try to help you to identify other things you might do instead of smoking.

What is your personal goal until our next call? Think of this as "tiny habits" and pair with something you do each day (e.g., When I brush my teeth, I will do two sit-ups.) Do you know which topic you'd like to discuss next time?

Document in Documentation Booklet

What would be the best date and time to call for that session?

Document in Documentation Booklet

Could you also verify the phone number to call?

Document in Documentation Booklet

Thank you. Do you have any questions for me before we end our call? I look forward to speaking with you again soon.

# **Rapport-Building**

Begin by asking the participant how she and the baby are doing.

#### **Documentation**

Go to the Documentation Booklet to complete initial questions. Based on responses, choose a topic theme to discuss from the list. If the participant is still smoking at all, continue with topic 4. If it is unclear which topic to proceed with, you may ask the participant which may be most helpful for her at this time.

Coaches Notes: This call is not intended to be a lecture, but to work with your client to come up with a way to deal with her daily stressors. It will work best if you actively engage her in discussion around her specific stressors and use this booklet for additional ideas on how she might deal with them. There is no need to review stressors the client doesn't mention.

#### **MANAGING DAY-TO-DAY STRESS**

Many people smoke because they believe it relieves stress, when the truth is that the only stress that is relieved from smoking is the stress from being a smoker (because it is only the withdrawal symptoms from smoking that are being addressed). Unfortunately, a lot of stress is unavoidable; however, the way we react to and manage stress can be controlled. This program will help you establish new ways to handle stress and not depend on tobacco.

We'll talk about some common stressors as well as some techniques for managing the stress without smoking. If you have your Healthy Mom, Healthy Baby Guide, it contains some ideas in this area and we'll be talking about some of them today.

# What are the main stressors in your life?

Document in Documentation Booklet and proceed to section that outlines participant's specific stressors to cover "Steps for Change." Review these Steps and ask participants if it feels like something they could do or if there are other things they can think of that would help.

## SPOUSE/PARTNER

When preparing to give up smoking, it's important to get your partner involved in the process. Whether your partner smokes or not, quitting is a big shift in your lifestyle and it's important that your partner supports you in the changes necessary to quit smoking.

## **COMMON SCENARIOS:**

Arguments or tense topics of conversation with your partner

- Feeling that your partner is trying to sabotage your goal to quit
- Financial stress caused by your partner or you
- Inability to communicate and be heard on things that are bothering you
- Not feeling connected due to stress

#### STEPS FOR CHANGE:

**Put it in writing**: Sometimes it's hard to express ourselves, and situations quickly get out of hand, but writing out the issues, your goals, and how the two of you could work together may be helpful.

**Prioritize time together**: It's amazing how beneficial some quality time together can be for a relationship. Plan things outside of your weekly routines and schedule regular times to do fun things together.

# **CHILDREN**

Coping with the demands on parents today is extremely tough, especially if you don't have a strong support system around you. However, there are ways to increase your support, prioritize family time, and decrease the stress.

#### **COMMON SCENARIOS:**

- Feeling overwhelmed by the demands of a new baby
- Feeling that you're not able to be there for your child as much as you'd like or they need due to work.
- Being overwhelmed by your children's schedules, i.e., team sports, clubs, school, driving them to and from appointments, etc.
- Behavioral issues or children that have special needs
- Custody issues due to a divorce

#### STEPS FOR CHANGE:

**Schedule in "you" time:** Taking time for yourself away from your new baby is important in recharging your battery. Even if it's a 15-minute shower during naptime or reading a magazine while your partner cares for the baby can help ease the stress of feeling needed all the time.

**Schedule additional time just with your children:** Spending just a couple hours together and making those hours fully focused on your time together will greatly benefit you and your children. Find a day of the week and avoid scheduling other things during that time.

**Make a shift in your routine:** Many family members come home and go to separate rooms watching TV, playing video games, etc. Make an effort to spend time together in the evenings, having dinner together, playing a game, or just talking and catching up on the day. Try turning the TV off and taking time with each other.

**Surround yourself with support**: Sometimes it's just not possible to do everything on our own and we need help from family and friends. Don't be afraid to ask for help, especially if it can benefit you and your children.

**Pool all of your resources:** In the case of custody issues or children with special needs, you may need to access different kinds of support. Be active in your child's educational plan, contact a mediator, and access assistance from social services or your employee assistance program. Start somewhere and even if you contact an agency that doesn't exactly offer what you need, chances are you will be directed to the right place.

# **WORK**

For many people, work can seem to take over our lives especially if you have a long commute to and from work and a demanding, high-stress job. Although work stress is certainly unavoidable a lot of the time, there are some ways you can become more efficient and less stressed during your day.

#### **COMMON SCENARIOS:**

- You feel underpaid for the work you do
- Your manager or co-workers are difficult to deal with
- The workload is overwhelming and never seems to lessen
- A long commute filled with traffic

#### STEPS FOR CHANGE:

**Tackle your day from a different angle:** If you're feeling overwhelmed, try to prioritize your day and make a list of tasks to be accomplished each day. It feels good to check off the list and see that you actually did get a lot accomplished for the day.

**Talk with your manager or supervisors:** You'd be amazed at some of the issues that can be dealt with by discussing your concerns with your manager or supervisor and asking for help.

**Carpool or Public Transportation:** Many people live far from work and are vulnerable to tobacco, as driving is a common trigger time. If you have the option, drive with others who don't smoke or take public transportation. These changes can help you cut down on tobacco, and save time and money.

**Look for a change:** If your job is having an overwhelmingly negative impact on your life, it may be necessary to explore your options for change.

#### **FRIENDS**

They are there when you need someone to talk to, relax and have a good time with, but if they don't respect your decision to quit, friends can also make your road to becoming free of tobacco that much more challenging.

#### **COMMON SCENARIOS:**

- You tend to meet up with friends at a bar or restaurant where you usually drink and smoke
- When friends come over or you go to their house, they still smoke in front of you or use tobacco
- Your friends don't want you to quit and may sabotage your attempts because they don't want to quit.

#### STEPS FOR CHANGE:

**Take a brief break:** You may have to spend less time with some of your friends and avoid socializing in typical places with them where you would usually use tobacco. This is only necessary until you're comfortable being around the tobacco without using it.

**Talk with your friends:** Discuss your plans for quitting tobacco and explain to them why you've decided to quit. If they understand that you're committed to quitting and would appreciate their support, they may be more likely to respect your decision. Ask your friends to join you in new activities that don't trigger your desire for tobacco.

**Spend more time with tobacco-free friends and family:** They will surely be an excellent support for you during your preparation to quit and staying tobacco-free.

# **FINANCES**

There are few people who are not impacted by the stress of money and finances. Today we have many additional costs including cell phones, cable and internet bills, higher gas prices, increased food costs, and more. With money, there never seems to be enough but as with any other stress contributor, there are ways to manage.

## **COMMON SCENARIOS:**

- You're hit with an unexpected bill during the month such as for unexpected medical needs or car repairs
- Feeling overwhelmed with credit debt and bills
- Never being able to catch up
- You are on a very tight budget
- Your partner poorly manages joint finances
- You spend more money on cigarettes per year and may pay more for life insurance and health insurance

#### STEPS FOR CHANGE:

**Re-evaluate/create your budget:** Sit down and look at what you're spending versus what you're making. Write down all of your expenses. There might be some necessary cuts to be made with your spending.

**Eliminate unnecessary spending:** Before you purchase something or commit to another bill, ask yourself, do you *need* this or do you *want* this? If it comes down to simply wanting, you can probably do without.

**Keep track of spending:** It's similar to when you go on a diet and count calories; it's amazing how those calories add up just as it is unbelievable how quickly we spend money without even realizing it.

**Get on the same page with your partner:** If one of you is in charge of the money, it's important for you both to be familiar with your budget and the status of your money.

**Advice from a financial advisor:** Again, if you feel that you're in over your head and not sure where to start to get back on track financially, you may want to sit down with a professional to develop a plan.

Determine how much money you will save from quitting smoking: Let's have a look at how much you will save when you're free of tobacco.

Help participant calculate savings in Documentation Booklet.

#### TIME MANAGEMENT

Juggling work, school, kids, family, and more is no easy task. We all need to step back sometimes and re-evaluate how our days and weeks are managed and see what we can do to save some time and sanity.

#### **COMMON SCENARIOS:**

- Work takes up most of your day and you have no time for yourself or family
- You've stopped taking care of yourself and spend most of your time taking care of others including, spouse, kids, parents, etc.
- You travel for work and have a schedule that often varies
- Over-committing and lacking the ability to prioritize daily tasks

#### STEPS FOR CHANGE:

**Keep a planner:** The more you can plan ahead, the better off you'll be. Each day, focus on tackling one thing at a time. This will also help you to avoid doubling up on appointments and spreading yourself too thin.

**Schedule in 'you' time:** It is essential to have personal time away from work, friends, family, appointments, and kids. If you've got a full schedule, see what

you can eliminate from your week and pencil in one hour a day or even a couple hours a week to focus simply on you.

**Learn to say NO:** Some people thrive on filling their days with commitments from sunrise to sunset. This can sometimes be detrimental to our health, to our families, and to our jobs. When you take time to breathe and have some down time, things may not seem so overwhelming.

# **HEALTH**

Most people who use tobacco understand the impact it has on their health. Unfortunately, many unhealthy habits come in pairs or even groups. You may not be getting as much exercise as you should, may have an unhealthy diet, drink more alcohol than is recommended, and neglect managing stress, as you rely on tobacco for that. When you combine all these unhealthy habits or even just a couple of them, your risk for many preventable diseases increases greatly.

#### **COMMON SCENARIOS:**

- You're limited in your ability to exercise due to your smoking
- You've been diagnosed with high blood pressure and tobacco is the main contributor
- You feel you've used tobacco so long that your health conditions are irreversible
- You're concerned about secondhand smoke and your family's health

#### **STEPS FOR CHANGE:**

*Understand the benefits to your health being tobacco-free:* Although *y*ou may have been using tobacco for 30 years, over time when you're tobacco-free, your body will recover and you'll feel the effects almost immediately.

**Work on implementing healthy habits to replace the tobacco:** Replace tobacco breaks with walk breaks. By eliminating a couple of the tobacco breaks during your work day, you may get more accomplished and feel less overwhelmed and stressed at the end of the day.

**Talk with your doctor:** Together with your doctor, you can create an appropriate diet and exercise plan to get you started.

#### LIFE CHANGES

Events happen in our lives that change things both positively and negatively. Because life is unpredictable, and due to the presence of the other stressors we discussed in this module, it can seem overwhelming to cope when a life change is added to the mix. Tobacco users, including those who have successfully quit, are at risk for relapsing or increasing their tobacco use during these times.

#### **COMMON SCENARIOS:**

- Positive stressors: switching jobs, buying a house, the birth of a baby, retirement
- Negative stressors: the death of a friend or family member, children growing up and moving away, divorce, a good friend relocating

#### SUPPORT DURING TIMES OF CHANGE:

**Surround yourself with friends and family:** It's always more difficult to deal with changes alone. Be sure to talk with your friends and family even if you can only reach them by phone.

**Seek out support groups:** There are always people in your similar situation that can relate to your experience. Whether it's a local support group in your community, online chat groups, or starting your own, sharing your feelings with others can be powerfully healing.

## **EMOTIONAL ISSUES**

If you've dealt with depression or anxiety in the past, you may experience similar feelings when quitting. As a result, it may be necessary to seek the help of a professional therapist that specializes in these matters. However, many of the stress factors we've discussed in this module can contribute to anxiety and depression. By taking a look at stresses in your life, establishing which ones play the biggest role in your emotional issues, and working with a professional, you can significantly reduce the impact they have on your life. Always contact your health care provider or therapist if you feel that your anxiety or depression is interfering with your daily life (e.g., sleeping, eating working).

**Action Plan:** Write down the stressors you experience each day over the next two weeks in your Healthy Mom, Healthy Baby Guide. Make a note of which ones trigger your desire to smoke.

What is your personal goal until our next call? Do you know which topic you'd like to discuss next time?

Document in Documentation Booklet

Please remember that any time you have the urge to smoke or are craving a cigarette, you can call our toll-free number 24 hours a day and someone will be available to talk with you about your cravings and try to help you to identify other things you might do instead of smoking.

What would be the best date and time to call for that session?

Document in Documentation Booklet

Could you also verify the phone number to call?

Document in Documentation Booklet

| Thank you. Do you have any questions for me before we end our call? I look |
|----------------------------------------------------------------------------|
| forward to speaking with you again soon. |

# **Rapport-Building**

Begin by asking the participant how she and the baby are doing.

#### Documentation

Go to the Documentation Booklet to complete initial questions. Based on responses, choose a topic theme to discuss from the list. If the participant is still smoking at all, continue with topic 5. If it is unclear which topic to proceed with, you may ask the participant which may be most helpful for her at this time.

Coaches Notes: You will likely know prior to this call whether or not the participant is partnered, but it is important to determine with certainty prior to the start of this call. If the participant is not currently romantically partnered, try to identify a household member or other support person for which this discussion will be relevant. For the purposes of this call, a partner can be a husband, wife, boyfriend, girlfriend, family member, friend, or any other person close to the participant.

# PARTNER SUPPORT

In this call, we'll be talking about how you can communicate with your partner to get the support you need while you're trying to quit smoking and stay quit. It isn't easy to quit smoking and stay quit, and it's important that you have a strong support system around you that will encourage you and keep you on track towards your goals. We've devoted a whole section to partners because we know that a person is more likely to quit smoking when they have strong partner support, and more likely to return to smoking if their partner smokes.

**Does your partner smoke?** (continue to box based on participant answer)

If yes, has this made quitting more difficult for you?

Document in Documentation Booklet

Stress levels are very high after a new baby joins the family, for both you and your partner. If your partner is a smoker, it may make it even more difficult if you see him/her dealing with a stressful situation by smoking when you're trying to quit.

You may want to **ask your partner to quit smoking with you**, as this would probably be the most supportive thing your partner can do as you try to quit. You can encourage each other through the hard times and remind each other why it's important to quit. You may want to share with your partner your reasons for wanting to quit and why a smoke-free household is important for the health of the baby as well as for the health of your family.

If your partner is unwilling to quit, **ask your partner to maintain smoke-free zones** in your home, your car, and in other areas where the baby will be. It will

be helpful to you if you don't see your partner smoking or smell the smoke, as this might tempt you to return to smoking. You might also ask your partner to hide any evidence of smoking in the house, such as ashtrays, cigarettes, or lighters.

Are you willing to talk with your partner about quitting or maintaining smoke-free zones?

Document in Documentation Booklet

If no, do you feel that this will make it easier for you to quit/stay quit?

Document in Documentation Booklet

Although it's great that your partner doesn't smoke, he/she can still trigger the desire to smoke again by not offering the support you need. For example, your partner may say things like "You were easier to deal with when you smoked" or "You're not eating for two anymore." Have an honest conversation with your partner about your need to hear kind words during this time and avoid teasing you.

#### Communication

It is very important that your partner is aware of your desire to quit smoking, your reasons for wanting to quit, and how he/she can help you on your journey to quit and stay quit.

Does your partner know that you (are trying to quit/quit) smoking?

If yes, what was your partner's reaction?

Have you felt supported by your partner?

If no, would you be willing to talk with your partner about this?

What do you think will be the hardest part of talking with your partner about your decision to quit smoking?

Document in Documentation Booklet

It may be helpful to make a list of all the ways you feel your partner can be the most supportive in your journey to quit smoking and share this list as part of your continuing conversation.

Possible ways your partner may support you (adapted from *Forever Free for Baby & Me*):

- By helping keep stress down (e.g., taking on more responsibilities in the home; exercising with you; playing with baby so you can rest)
- By celebrating successes (e.g., cooking you dinner when you complete an action plan in the program or don't smoke when you normally would; offering compliments about how nice you smell)
- By providing practical support (e.g., bringing home your favorite gum to chew instead of smoking)
- By asking how to help
- By being patient, supportive, and listening
- By not expecting overnight success

As part of the conversation, it is also important that you understand how your quitting smoking may impact your partner.

# How might your partner be impacted by your quitting smoking? Document in Documentation Booklet

Examples of ways your partner may be affected by your quitting smoking (adapted from *Forever Free for Baby & Me*):

- Loss of a smoking partner (if he/she smokes)
- Increased sense of responsibility to help you quit
- Coping with possible withdrawal symptoms you may face (e.g., irritability)

**Action Plan:** Have a conversation with your partner about how he/she can best support you on your journey to quit smoking or stay quit.

What is your personal goal until our next call? Do you know which topic you'd like to discuss next time?

Document in Documentation Booklet

Please remember that any time you have the urge to smoke or are craving a cigarette, you can call our toll-free number 24 hours a day 7 days a week and someone will be available to talk with you about your cravings and try to help you to identify other things you might do instead of smoking.

What would be the best date and time to call for that session?

Document in Documentation Booklet

Could you also verify the phone number to call?

Document in Documentation Booklet

Thank you. Do you have any questions for me before we end our call? I look forward to speaking with you again soon.

### Rapport-Building

Begin by asking the participant how she and the baby are doing.

#### Documentation

Go to the Documentation Booklet to complete initial questions. Based on responses, choose a topic theme to discuss from the list. If the participant is still smoking at all, continue with topic 6. If it is unclear which topic to proceed with, you may ask the participant which may be most helpful for her at this time.

Coaches Notes: Regardless of how long your client has been a tobacco user, she has undoubtedly integrated this addiction into her daily life. She has established systems to ensure that she has access to her tobacco at regular intervals throughout the day and may have created a support network of other tobacco users. Asking your client to remove all of these rituals from her daily life without replacing them with alternatives is not a good way to ensure success. Use this call to discuss common hurdles that are faced when someone quits using tobacco and discuss steps to take to remove these barriers from her ability to quit. Ask your client to open her Healthy Mom, Healthy Baby Guide to this topic so that she may follow along with you.

### **Breaking down Common Barriers**

This call will review some of the everyday barriers and challenges that may arise when quitting tobacco and how to overcome them.

Despite the health consequences, when listing the pros and cons of tobacco use, most people have a few pros such as, "I like tobacco" or "I love a cigarette with my coffee or after a meal". Of course there are perceived benefits from smoking; otherwise people wouldn't do it. However the negative side of the list greatly outweighs the positive.

What are the benefits you get from smoking and how might you prepare yourself to break through this barrier to quitting/staying quit?

Document in Documentation Booklet and proceed to section that outlines participant's specific benefits from smoking to cover "Preparing to Quit" section.

Let's talk about the ones you mentioned. In your Healthy Mom, Healthy Baby Guide are several common barriers people are faced with when trying to quit tobacco, along with ways to break through the barriers that you can also reference.

## \*Tobacco is one of My Best Friends

You turn to tobacco during a stressful day or when you're just home alone. It's been good company but now it's time for you to look into other forms of support because with friends like these, who needs enemies? **Talk with your family, friends, and co-workers to let them know you're serious about quitting and would appreciate their support.** The more people you can surround yourself with the better.

**Preparing to quit:** Let your co-workers, friends, and family know that you are quitting tobacco so that you can build your own support group and have people to talk to when the process gets tough.

### \*Tobacco is a Huge Part of My Day

For many people, common triggers to use tobacco include a break at work, after a meal, talking on the phone, driving in the car, etc. Through this program and developing your quit plan, it's vital that you work to change your daily routines so that you're able to avoid those common trigger times and replace them with alternative actions. For example, if you spend a lot of time on the phone and find that you smoke; give yourself a time limit to spend talking, such as 5 minutes so you won't be inclined to reach for a cigarette or make your calls from a place you cannot smoke.

**Preparing to quit:** Look at the common times you smoke throughout the day and think about some alternative things you can do instead. Start with just one time each day and use that opportunity to do something positive instead of smoking.

\*Smoking Calms me down when I'm Feeling Stressed or Anxious
For those who have been smoking almost their entire lives, their ability to handle
stressful situations without tobacco is greatly impaired. As part of your plan to
quit tobacco, it's essential that you explore alternative ways to manage
your stress and anxiety. There are many ways to reduce stress with relaxation
techniques, exercise, talking with supportive friends and family, reaching out to
your health counselorand looking at your lifestyle to see how you can reduce
some of the factors contributing to the stress and anxiety.

Preparing to quit: What have you done in the past during times of stress without smoking? Can you reduce stress in your life so that you're not so dependent on tobacco to get you through the daily stressors? What little change could help? This may take some examination of the bigger picture to see what is contributing to stress in your life and if there are things you can do to enact a positive change.

\*Smoking Allows an Opportunity to Step Away from Work and Stress

Imagine how much more productive you could be with your day or the positive things you could be doing with that time you spend smoking. For people who claim they have no time, try adding up the time you spend centering your day on smoking. A few 5-10 minute smoke breaks throughout the day, in the morning before work, and the evenings after work really add up.

**Preparing to quit**: Calculate a rough estimate of the amount of time you spend smoking in any given day. What are some other ways you might spend that time? One option might be spending more time with your baby: reading, going for stroller rides, or playing with him/her.

## \*Smoking Keeps me Occupied

Have you noticed you smoke less when you're working or busy with projects at home? While trying to quit, it's important to fill up the down time at home on the weekends or in the evenings with tasks or things you've wanted to accomplish but may be putting off. Many people tend to use tobacco more in the evenings and on the weekends when they don't have work to keep them busy.

**Preparing to quit:** It's likely that the new baby is keeping you very occupied, but if you find that you have down time, make a list of projects you have wanted to start, hobbies you've been interested in trying out, or other goals you've wanted to focus on. Think about how you will feel when you start crossing completed items off of your list. Try to focus on small changes.

## \*Smoking Helps me Eat Less

Many people avoid quitting tobacco because nicotine acts as an appetite suppressant. It's important to tackle one thing at a time. First, focus on developing a plan to quit tobacco. Setting small, attainable health goals to improve eating habits or increase exercise can actually help you cut down on cigarettes (e.g., I will eat at least one serving of fruit with each meal). Much of what we discuss in this program is about replacing the unhealthy habits with positive, healthy ones.

Preparing to quit: Take advantage of opportunities to make more time for your health in place of a few cigarettes throughout your day. For example, instead of reaching for a cigarette first thing in the morning, make yourself a healthy breakfast, play with your baby, or take a short walk. Make one of your usual smoke breaks a walking break or take your baby out for a stroller ride. These examples will not only get you smoking less but will help relieve stress and improve your overall health. Take it one cigarette at a time.

It is important to identify your personal barriers so they can be accounted for in your quit plan and approach. Otherwise you run the risk of being tripped up by them and experiencing a set back.

**Action Plan:** If you think of any additional barriers to quitting smoking/staying quit over the next few weeks, write them in your Healthy Mom, Healthy Baby Guide and make a plan for how you might overcome these.

What is your personal goal until our next call?

Document in Documentation Booklet

Please remember that any time you have the urge to smoke or are craving a cigarette, you can call our toll-free number 24 hours a day 7 days a week and someone will be available to talk with you about your cravings and try to help you to identify other things you might do instead of smoking.

What would be the best date and time to call for that session?

Document in Documentation Booklet

Could you also verify the phone number to call?

Document in Documentation Booklet

Thank you. Do you have any questions for me before we end our call? I look forward to speaking with you again soon.

## Rapport-Building

Begin by asking the participant how she and the baby are doing.

### Documentation

Go to the Documentation Booklet to complete initial questions. Based on responses, choose a topic theme to discuss from the list. If the participant is still smoking at all, continue with topic 7. If it is unclear which topic to proceed with, you may ask the participant which may be most helpful for her at this time.

Coaches Notes: This week is very important in the development of a unique quit plan for each of your clients. This call will help your client think through all aspects of her quit plan and compile her ideas and strategies into one document. Encourage your client to share her quit plan with family, friends, and colleagues who will support her in her process. Encourage her to include as much detail as possible in her plan... a strong foundation in this area will help her to navigate the challenges and hurdles she will face as she breaks this addiction.

## THE QUIT PLAN

In this call, you will have the opportunity to develop your personal quit plan that you can easily reference throughout your journey to quit smoking and stay quit.

In the previous weeks, this program provided you with ideas and information on some of the tools needed to develop a personalized quit plan that works for you. Being prepared is the key to beginning a tobacco-free life. In this section you will make a plan of action for quitting. With a solid and well thought-out plan, you will be equipped to overcome obstacles that may arise during the quit process. Your personal quit plan will consist of the following:

- Understanding why you smoke
- Identifying your reasons for wanting to guit
- · Identifying people who will support you
- Recognizing triggers and how to overcome them
- Thinking about support methods, such as nicotine replacement therapy
- Choosing a quit date
- Exploring whether you want to guit all at once or cut back to get ready to guit

## **Understanding Why You Use Tobacco**

We all know that using tobacco has negative health effects. So why do so many people keep using it? Nicotine is an addictive substance, like alcohol or drugs, which keeps people dependent upon the soothing effects they receive after smoking or using other types of tobacco. Just like any addiction, there are three

components that need to be addressed in order to successfully quit. Let's look at each of these three areas in detail and determine where you will need to focus your efforts.

**#1 Physical Addiction to Nicotine:** Nicotine is an addictive substance that causes changes in the brain that make you want to use it more and more. When your body does not have nicotine, there may be unpleasant feelings and cravings. However, when you get nicotine again, the good feelings come back and the craving goes away. So, one part of quitting is realizing there is a true physical addiction to nicotine and planning ways to overcome the possible withdrawal symptoms. Common withdrawal symptoms include difficulty sleeping, increased appetite, restlessness, difficulty concentrating, irritability, a depressed mood, or anxiety. The good news is these feelings will not last forever!

Not everyone will have symptoms when they stop using tobacco, but the longer you have used tobacco and the more frequently you've used it increase the likelihood that you might experience withdrawal. Typically, once you quit using tobacco, it takes about 6-8 hours for the nicotine to leave your body and withdrawal can start within a few hours of your last use. The unpleasant side effects of not having nicotine peak within 1-4 days after quitting and might last for up to 1 or 2 weeks (though for some may last longer).

## Are you physically addicted to nicotine?

Document in Documentation Booklet

If you answer "yes" to two or more of the following you may be addicted to nicotine. Circle your answers:

- 1. Do you need to have a cigarette first thing in the morning?
- 2. Do you smoke one pack (20) of cigarettes or more a day?
- 3. When you cannot use nicotine, do you feel a craving for it?
- 4. When you are sick enough to stay home from work in bed do you still smoke?
- 5. Do you ever feel like you "need" to have a cigarette?
- 6. Have you ever tried to quit tobacco before and failed?

**#2 Psychological Dependence:** While the withdrawal symptoms you might experience after quitting tobacco will go away after your body has been weaned from nicotine, the psychological dependence is a more lingering challenge that needs to be addressed. The psychological components of tobacco use are the emotional reasons that you smoke. Some people smoke to cope when they feel

emotions like stress, anxiety, boredom, or other feelings that they might have difficulty handling otherwise. Smoking also tends to be psychologically connected with positive emotions and experiences like celebrations and spending time with certain friends and family.

In some ways, you may have thought that nicotine is your best friend. You have used it through many emotional situations and everyday occurrences. However, this is a "friend" who can kill you! In order to be a successful quitter for the long haul, it is important to learn new and healthy ways to deal with your emotions.

Identifying the emotions that may contribute to your dependence on nicotine will provide you with more useful information to help you create a solid quit plan. Take a look at the list of feelings below and circle the emotions that you cope with by using tobacco. List any others that are relevant for you in the blank spaces.

| Anger | Stressed at work | Нарру |
|-----------------------|------------------|---------|
| Sadness | Tired | Boredom |
| Stress about finances | Hunger | Excited |
| Stressed at home | Unsure | Nervous |

#3 The Routine of Tobacco Use: One of the more difficult parts of quitting tobacco is overcoming the routine of smoking. Using tobacco often becomes a part of our everyday routine whenever we have spare time to fill. For example, whenever you finish a meal or get in your car, you automatically have a cigarette. When tobacco use becomes routine, you are no longer making a conscious choice to smoke.

The most common strategy that people use to break the routine of tobacco use is willpower. But willpower alone is not a long-term solution!!! You may have noticed this fact if you have tried to quit before or if you have tried to make other lifestyle changes such as losing weight or starting an exercise routine. You were probably successful for a couple of days and then went back to your old ways.

Fortunately, there is another path to take:

Identify your current routines related to tobacco use and create new routines that support your long-term goal of being tobacco-free. For example, instead of having a cigarette after a meal, you may choose to take your baby on a stroller ride around the block. Or on your drive home, you might try listening to audio books on your car stereo.

Now, let's take a look at your routines related to smoking to pinpoint areas for possible change. This exercise is important for increasing your awareness of your tobacco use. Once you are aware of what your routines are, it is easier to create new routines to take the place of the old ones.

Place a check mark in the box next to the situations when you typically smoke or use other forms of tobacco. Feel free to add your own in the blank spaces. Make note of the top three that stand out the most.

| ☐ After finishing a meal | ☐ While driving in my car |
|---|---|
| ☐ While taking a break with co-workers | ☐ With an alcoholic beverage |
| ☐ With a cup of coffee | ☐ While talking on the telephone |
| ☐ When putting off a project | $\hfill\square$ When around other smokers |

## **Triggers**

Identifying your personal cues or signals that lead to tobacco use is a crucial step in developing your quit plan. Triggers are actions that make you want to use tobacco, such as seeing someone else smoking, driving in your car, social gatherings, a certain time of the day, stress, smelling cigarette smoke, difficult emotions, certain beverages, etc. These triggers result in urges to use tobacco. For example, you get into your car to drive to work and as soon as you get on the road, you light up a cigarette. You've connected driving in the car with smoking; therefore driving is your trigger. By identifying your unique cues, you can find alternative activities and thoughts to replace using tobacco. Easier said than done, right? Yes...changing any behavior is challenging. However, with a clear plan of action, you can be successful! Our main goal is to break the association that you have between using tobacco and what you normally do or think, and this task is accomplished by increasing your awareness.

Take some time to write down common actions, thoughts, or feelings that you associate with the urge to smoke. Make sure you create a list ahead of time because if you wait until the urge occurs to try and come up with an alternative, the chances of not smoking are not as high.

| <u>Trigger/Thought</u> | Alternative Action/Thought |
|---------------------------|-------------------------------------|
| Drinking coffee | Drink tea instead of coffee |
| I really need a cigarette | Smoking isn't a need, it is a habit |
| | - |
| - | |
| - | |

### **Reasons for Quitting**

Everyone has a different reason for embarking on the quit tobacco journey. You may want to quit solely for the health of your baby, to improve your own health, or to save money. You may be motivated to quit for the benefit of your family or friends. Maybe you are concerned about the effects of secondhand smoke on your family, or perhaps your loved ones are concerned about your health. Whatever your reasons for quitting might be, having a list that you can refer back to can be helpful during challenging times. Why do you really want to quit smoking? Write down the reasons and benefits you come up with below. No reason is too big or too small and there are no wrong answers.

| I want to stop smoking because (include financial, health, social, etc. reasons |
|---|
| I will benefit from quitting because: |
| My baby will also benefit because: |
| It also important to consider why you may <b>NOT</b> want to quit. Quitting something that is such a large part of your everyday life can be scary and overwhelming. |
| I don't want to quit because: |

When you are finished with this section, be sure to choose the reasons and benefits that mean the most to you and write them in your quit plan.

### Personal Support

Quitting tobacco is not easy, so the more support you have the better. Support can come from family, friends, co-workers, online communities, or tobacco cessation programs. You will most likely find that people are very supportive of you quitting smoking. Be sure to surround yourself with these people as much as possible during the quitting process and reach out to them

instead of tobacco if you are in need of help. If possible, try to find a friend or partner who also wants to quit and do it together. Going through the process with someone else can help during challenging times.

Think of people, programs, websites, etc. that you can rely on during your quitting process. Who/what will be helpful and why?

Helpful people:

Websites, support groups, and cessation programs I may use are:

### **Baltimore Resources**

- Freedom From Smoking® Class this free seven week program uses a positive behavior change approach, and helps participants develop their own plan on how to quit. In eight 90-minute sessions, you'll learn about reducing stress, cravings, and withdrawal symptoms, and how to control your weight while resisting the urge to smoke. To get information on when the next session starts, call 410-887-3828.
- Tobacco use Prevention and Cessation Program call 410-887-3828 to speak with a staff member. They offer free nicotine replacement gum, lozenges, smoking cessation classes and support.
- Baltimore City Health Department provides free smoking cessation group therapy and patch therapy
- **Good Samaritan Hospital** offers a smoking cessation support group that meets weekly, Mondays 6:30pm-8pm
- women.smokefree.gov

### Medications

Having support in the form of nicotine replacement therapy (NRT) or alternative approaches can be invaluable in helping you quit. It is always important to discuss these options with your health care provider before making any final decisions. Be sure to review the section in your Healthy Mom, Healthy Baby Guide on nicotine replacement therapy and alternative approaches to decide which options are right for you. Since some NRTs and medications take time to get and may require you to talk with your doctor, it is necessary to plan ahead.

| I have used the following NRT or medications in the pathem again: | in the past and p | past and plan on using |
|---|---|---|

| I have used the following NRT or medications in the past but they did not work well for me because: |
|---|
| I plan on trying NRT or medications again but changing the way I use them by: |
| I also want to try the following alternate support methods (e.g., meditation, acupuncture, relaxation exercises) and think they will be helpful because: |

### **Your Quit date**

One of the first steps to take when quitting tobacco is establishing a quit date. The quit date is the day you will become a non-smoker! It's important not to put off this date. Is there a significant day, such as a birthday or anniversary, coming up within the next 2 weeks that you want to quit by? Once you pick a date, make sure it is at a time that is convenient for you and that is not stress-laden (i.e., the holiday season). And remember there are no time limits. You can set your quit date for two days from today or two weeks. After you have selected your quit date, be sure to make note of this special day in a visible place! It marks the beginning of your life as a non-smoker or the beginning of a tobacco-free life. You may choose to start letting important people in your life know about your plans and telling them how they can best support your efforts.

# Do you have a date in mind for your Quit Date?

Document in Documentation Booklet

Coaches Notes: It is critical to check in with your client on her Quit Day. Your client may find that certain aspects of her plan are not working and may need your assistance to make adjustments. Encourage your client to reward her success.

### **Quitting all at once vs. Cutting Back**

Which is the best way to quit? All at once, or by slowly tapering down your tobacco use? As we discussed before, quitting smoking involves not only ridding your body of nicotine, but also changing behaviors. Because changing behaviors takes time, the most effective way to quit tobacco is to slowly cut back while

forming new habits and making sustainable behavior changes. It also helps to gradually wean your body from the nicotine it has been used to so withdrawal symptoms are minimized.

Sometimes we decide that we really want to quit TODAY and we forge ahead cold turkey without a solid plan in place. In this case, we are relying on willpower and willpower does not work for long. Whether you decide that you want to quit all at once or to gradually cut back, be sure to weigh all of your support and NRT/medication options and create a plan to quit. Taking these steps will greatly increase your chances of long-term success!

# Decide which method will work best for you by answering the following questions:

How have you tried to quit in the past? If so, which method did you use at that time? What worked about that method and what didn't work? Which method do you think will be most effective for you now and why?

**Action Plan:** Complete your Quit Plan this week and share it with any friends and family who are willing to support you in your quit. I'll also give you a call on your quit date just to check in.

What is your personal goal until our next call? Do you know which topic you'd like to discuss next time?

Document in Documentation Booklet

Please remember that any time you have the urge to smoke or are craving a cigarette, you can call our toll-free number 24 hours a day 7 days a week and someone will be available to talk with you about your cravings and try to help you to identify other things you might do instead of smoking.

What would be the best date and time to call for that session?

Document in Documentation Booklet

Could you also verify the phone number to call?

Document in Documentation Booklet

Thank you. Do you have any questions for me before we end our call? I look forward to speaking with you again soon.

### Rapport-Building

Begin by asking the participant how she and the baby are doing.

### Documentation

Go to the Documentation Booklet to complete initial questions. Based on responses, choose a topic theme to discuss from the list. This is a good call to do after a person has created or reviewed a quit plan and quit smoking, but can be done towards the end of the PPCC program if other topics have been covered. If it is unclear which topic to proceed with, you may ask the participant which may be most helpful for her at this time.

Coaches Notes: Lapses and relapses are part of the process for many people trying to quit tobacco, and are especially common in the postpartum period. If your client returns to using tobacco products in any amount, you should take it seriously and should make significant attempts to reengage her in the process and encourage her that all is not lost. Many tobacco users will feel as though they have failed if they slip up once or twice, but you can help them to understand that they can learn from this experience and move on. Help them to analyze why they lapsed and put together an action plan to prevent it if they are in that situation again. Encourage your client to try many different strategies until she finds the one that works for her.

## **RELAPSE PREVENTION**

This call will discuss approaches for preventing a relapse or return to old smoking patterns. Common obstacles to staying quit are identified and tips to overcome them are given.

Chances are you've tried to quit tobacco in the past. Maybe you were successful for a day or even a year. If you've experienced a relapse in the past and feel that you've failed, don't worry, you're not the first or the last to return to old routines. The truth is it takes the average tobacco user more than a few tries to quit tobacco once and for all. The majority of people who quit go back to using tobacco, not because it is impossible to quit, but because they were unprepared. This call will help you avoid a relapse and overcome a slip.

### Lapse versus Relapse

A lapse is a slip, a mistake. It does not mean you have failed at being tobaccofree. A lapse often occurs when you are in a situation where you would have smoked in the past and don't quite have the tools to handle it. For instance, if you are stressed and go for the most familiar way to reduce your stress, smoking a cigarette, and realize afterwards what happened, that is considered a lapse. You realize what went wrong, come up with strategies to deal with the situation should it come up again, and get right back on track. It is normal and part of the quitting process to have one, or even a few, lapses.

A relapse is a series of events that causes you to fall back into an unhealthy way of life (i.e., a smoking addiction lifestyle), after a period of improvement. A lapse can easily become a relapse if you give up and go back to using tobacco. You are most vulnerable to a relapse during the time that you are withdrawing from nicotine and trying to solidify new behaviors, but a relapse can happen years down the road as well. **Awareness is key in preventing a return to tobacco use.** At some point you will probably notice your confidence rising and you will start to let your guard down a bit. That is when thoughts such as "just one cigarette won't hurt" can creep in and wreak havoc. However, there are steps you can take to stay tobacco free.

Here are some tips to overcoming slips:

## Tips to overcome a slip

- ✓ Don't wait to take action, a slip can easily lead to a relapse
- ✓ Stop using tobacco immediately and throw away all tobacco and related items
- ✓ Remove yourself from the situation that led you to using tobacco again.
- ✓ Evaluate what led to the slip: Where were you? Who were you with? What were you doing? How were you feeling?
- ✓ Review your personal quit plan for strategies to deal with triggers
- ✓ Call your Counselor or friends for personal support for encouragement

# Remember, you have not failed and you can overcome a slip! Don't give up!

The best way to prevent a relapse is to plan ahead and prevent one from occurring in the first place. Be aware of the following behaviors or attitudes that can make you more susceptible to relapsing:

- Being overly confident
  - Never underestimate the power of nicotine. When some people start feeling better, they develop a false sense of control over their addiction to nicotine. This attitude quickly leads to the belief that they can socially smoke or just have one cigarette.
- Expecting perfection
  - Just like other goals you have attempted to reach, quitting tobacco has peaks and valleys. Be gentle with yourself and practice positive self-talk when you veer off course. Keeping this point in mind is vital, especially if you experience weight gain or other things that you view as negative aspects of quitting smoking. Don't try and lose weight while you are

quitting. Things will return to a more balanced point and that is the best time to make other significant changes in your life.

- Underestimating the need to be adequately prepared with a quit plan
  - As the saying goes, "failing to plan is planning to fail". Adequate preparation is essential to long-term success. Keep in mind that you may need to make adjustments to your plan along the way.
- Rationalizing about the benefits of smoking when cravings appear
  - You might find yourself thinking "Smoking helps me focus so I perform better at work" or "I already cut back to a safe level so I don't need to quit". These thoughts are strong triggers to relapse and creating counter statements about the truth of the matter is a powerful antidote.
- Feeling overly stressed
  - You are more likely to relapse during times of high stress. Developing positive strategies to handle stress is critical to staying quit. Exercise, counseling, breathing exercises, and learning time management skills can all greatly improve your ability to cope.

### **Overcoming Obstacles**

In your personal quit plan, you had a chance to plan for challenges associated with quitting such as triggers, and in a previous call, we discussed common barriers to quitting. Be sure to review your quit plan to remind yourself of what you listed as your personal triggers and how you will overcome them. Here we will discuss in more detail some common triggers or situations that lead to a lapse and how to successfully deal with them.

**Triggers:** The longer you go without using tobacco, the easier it will be to overcome your triggers. This is partially due to a reduction in cravings for nicotine. At first you may need to separate yourself from certain situations, but as you get used to not using tobacco, you can slowly return to certain activities because the likelihood of feeling the urge to smoke is decreased. There may be certain activities that you won't return to but ultimately the choice is yours.

# What situations will be most difficult to face when you're not smoking? How will you deal with them?

Document in Documentation Booklet

**Stress**, anxiety and negative moods: One of the most common reasons that someone returns to using tobacco is stress. Nicotine tends to calm nerves and gives you a temporary feeling of being relaxed. Now that you are a non-tobacco user, you need to learn to deal with stress and negative moods without tobacco. When a negative event happens, you will at first have the urge to reach for tobacco in order to cope. It is the easiest solution because you have used it many times before; however, keep in mind that using tobacco will not cause the problem to go away.

**Excitement and positive moods:** Another common reason that people start using tobacco again is related to happy events in their life. Smoking in particular is a very social activity so it is a usual part of birthday parties and other types of festivities. Alcohol, which can be a major trigger for smoking, is frequently associated with celebrations, thus making it difficult to not smoke.

What moods have you found contribute to your desire to use tobacco?

What are new ways that you can use to improve your mood or to celebrate?

Document in Documentation Booklet

Alcohol/Bar scene: About half of the people who relapse do so because of an alcohol-related event. Our inhibitions and reasoning skills are affected after a few drinks, making it harder to resist tobacco. The quit plan pretty much goes out the window! Because tobacco is found at places where alcohol is served, such as bars, it is often best to avoid such establishments until you are sure of your ability to stay quit.

List 3 new ways that you can socialize with friends and loved ones that will support your goal of being tobacco-free.

Document in Documentation Booklet

Friends/family who smoke: Staying quit is often a challenge for people who live with or are around others who smoke. Certainly living with others who use tobacco presents a significant obstacle. Communication about your need to stay tobacco-free is essential to your long-term success. If the people you live with who smoke are not interested in quitting, the best thing to do is get their support to designate tobacco areas. For example, only allow tobacco use outside, be clear about no smoking in the house, and set some boundaries about leaving tobacco -related items lying around the house. You can talk about how the smoke affects not only you but the baby, and how important it is to maintain a smoke-free home for the health of the baby. Be clear that it is not ok for them to offer you cigarettes, even if you ask. You may need to make similar requests from co-workers or friends.

Who do you need to communicate with about your quit goals and what do you need to request?

Document in Documentation Booklet

**Tip to Quit:** Lapses may happen over the course of your quit. Recognize it, strategize for the future, and keep following your plan! This is the best way to prevent a lapse from becoming a relapse.

**Action Plan:** For each of the following scenarios, write how you would handle them without resorting to tobacco.

- 1. I can't stop thinking of using tobacco when I am taking care of the baby:
- 2. I am so stressed at work that I need to use tobacco to calm down:
- 3. I got a promotion at work and am so excited I want to celebrate with tobacco:
- 4. My friends are going out to our usual bar on Saturday night where there will be smoking:
- 5. My partner uses tobacco and it makes me want to use tobacco more:

What is your personal goal until our next call? Do you know which topic you'd like to discuss next time?

Document in Documentation Booklet

Please remember that any time you have the urge to smoke or are craving a cigarette, you can call our toll-free number 24 hours a day 7 days a week and someone will be available to talk with you about your cravings and try to help you to identify other things you might do instead of smoking.

What would be the best date and time to call for that session?

Document in Documentation Booklet

Could you also verify the phone number to call?

Document in Documentation Booklet

Thank you. Do you have any questions for me before we end our call? I look forward to speaking with you again soon.

### Rapport-Building

Begin by asking the participant how she and the baby are doing.

### **Documentation**

Go to the Documentation Booklet to complete initial questions. Based on responses, choose a topic theme to discuss from the list. This topic can be done at any time, but preferably after the woman has quit smoking. If it is unclear which topic to proceed with, you may ask the participant which may be most helpful for her at this time.

Coaches Notes: It is important to note that quitting tobacco is a significant behavior change that needs to be the sole focus for your client in the beginning weeks and months of her quit process. Often, clients want to work on other behavior changes simultaneously, such as weight management or increased physical fitness. This topic is designed to help your clients to maintain and even improve their overall health while they quit tobacco use, without detracting from their quit process. Weight gain is a common side effect with quitting tobacco and is a significant concern for some individuals. Encourage them to focus on healthy eating and moderate exercise while they quit tobacco and let them know that they can address any weight gain after they have fully completed their program.

## **Eating Well and Staying Healthy While Quitting Tobacco**

Taking care of yourself is a great strategy to help you stay quit, and is also important now that you have a new baby. This call will review basic nutrition and exercise guidelines and tips for losing any post-tobacco weight gain. It may also help you lose the "baby weight."

When you are trying to guit smoking, that effort should be your number one priority. However, you might be surprised to learn that healthy nutrition and exercise can support you in your goal to become tobacco-free. Short breaks for exercise can reduce cravings, and healthy snacks are a good way to occupy your mouth as you step away from smoking. If the weight gain that is common with quitting tobacco is a concern for you, good nutrition and exercise will help you to minimize it, and will allow you to stay focused on your number one goal.

### The Cause of Weight Gain and Increased Appetite

 Nicotine acts as an appetite suppressant. While using tobacco, your weight can drop due to reduced food consumption. When you guit, your appetite may increase and you may eat more as a result. You also may find that you replace some of your usual tobacco with food.

- The average weight gained as a result of quitting tobacco is 6-8 pounds.
   During the first week of not using tobacco, up to 3-5 pounds of weight gain may be due to water retention.
- Nicotine causes an increase in blood pressure, heart rate, and an increase in your metabolism. This means when you quit tobacco, your body may use fewer calories.
- Try to incorporate three small meals and two snacks into your day. This
  eating style will help keep your metabolic rate revved up to counteract the
  impact that nicotine would have had. And don't forget breakfast...it truly is the
  most important meal of the day! This is especially important if you are
  breastfeeding your baby.

**Put it to Action:** Allow yourself to fluctuate up to 10 pounds without panicking. The weight gain will only be temporary and you can focus on losing any additional weight after you're comfortably tobacco-free!

## **Substituting Tobacco with a Healthy, Delicious Snack**

- Right now you may feel that you don't have the time or energy to devote to healthy eating, but quitting tobacco requires a shift in priorities and some small alterations to your daily routines. Remember that you are saving time each day by not using tobacco, so try to use those extra minutes for healthy meal planning. This benefits not only you, but your baby if you are breastfeeding.
- Do celery and carrot sticks come to mind when you think of healthy snacks?
  The good news is that there are many other tasty and satisfying options to
  explore. Instead of reaching for junk foods, be sure to have some nutritious
  snack options on hand at work, at home, in the car, and in any other location
  where you spend time regularly.
- Don't wait until you are overly hungry to take the time to eat. If you go too long between meals, your blood sugar levels will drop and you will find it more difficult to control your food intake.

**Put it to Action:** In the morning or the night before work, pack 2-3 healthy snacks to bring with you during your day.

## **Increase your Physical Activity**

 Exercise has countless benefits, and when you are trying to quit tobacco, it can be a perfect distraction from cravings and a healthy replacement for smoking.

- Managing stress is essential when quitting tobacco. Exercise is one of the most effective ways to keep stress low while also improving your health.
- Studies have shown that people who incorporate 45 minutes of walking into their day gain less than 3 pounds when quitting (as compared to the average weight gain of 6-8 pounds).
- There are several simple ways to boost activity in your weekly routine such as taking the baby for a walk in the stroller, joining a gym, starting a walking program with other new moms, using home equipment, or finding a friend or family member to exercise with.

If you haven't been active recently, or if your doctor has not cleared you for exercise yet, please speak with your health care provider about when you may start any exercise program.

**Put it to Action:** If you have a tight schedule, break up the 45 minute time goal into three 15 minute walks during the day. For example, one walk with the baby in the morning, one during your lunch break, and one in the evening before or after dinner. Your baby will enjoy this time spent outdoors with you!

## Sleep, Hunger & Energy Levels

- Sleep is an important component of a healthy lifestyle. Without adequate sleep, you may not have enough energy for your daily tasks let alone exercise and resisting the urge to use tobacco.
- Studies have shown links between certain hormones that affect hunger levels influenced by lack of sleep.
- Getting a sufficient amount of sleep can boost your energy levels, which will help you to increase activity and make healthier food choices.

**Put it to Action:** It may be difficult to get more sleep with a new baby in the house. If you feel you could use more sleep, this week, try to nap when the baby naps and go to bed 30 minutes earlier than usual.

## **Balanced Daily Meal Plan**

If you're not sure what to eat or how to create a balanced diet that will give you sustained energy throughout the day, here is a simple breakdown:

• **Fruits and Vegetables:** Base your meals around seasonal produce. Fruits and vegetables are low in calories, rich in vitamins, minerals and fiber.

- Whole Grains: Choose whole grains such as wild rice, whole grain pastas, quinoa, whole grain couscous, brown rice, oatmeal, and barley. These grains contain more nutrients and fiber than their processed counterparts.
- Lean Proteins: Food proteins are the building blocks of body proteins and are an important component of a balanced diet. Choose lean protein sources such as chicken, turkey, and fish more often than beef and pork as they are excellent sources of protein with less cholesterol, saturated fat, and calories.
- Healthy Fats: Avoid saturated fats and cholesterol while getting
  monounsaturated and polyunsaturated fats from plant sources such as olive
  oil, canola oil, nuts, avocados and fish.
- **Fiber:** The recommended daily intake for fiber is at least 20 grams per day for women and at least 30 grams per day for men, yet on average, people get just 15 grams each day. By adding more fruits, vegetables, and whole grains to your diet, you will also be increasing your dietary fiber intake.

To simplify the amount of each of the above that you should eat, try thinking of it this way. Imagine you have a plate that is divided into four sections. One-half of the plate should be made up of fruits and vegetables, one-quarter of it should be a lean protein, and the final quarter should be a whole grain. Add a healthy fat and you are ready to eat!



### The Bottom Line

You are making a significant lifestyle change right now by becoming tobaccofree. And it is a great time to look at the other ways you can begin to live a healthier life. By replacing the unhealthy habits with healthy ones, you'll be more likely to have long-term success and reach your ultimate goal.

**Action Plan:** Choose one meal every day this week that matches the healthy plate model provided in this session. Remember, one-half of the plate should be made up of fruits and vegetables, one-quarter of it should be a lean protein, and the final quarter should be a whole grain.

What is your personal goal until our next call? Do you know which topic you'd like to discuss next time?

Document in Documentation Booklet

Please remember that any time you have the urge to smoke or are craving a cigarette, you can call our toll-free number 24 hours a day 7 days a week and someone will be available to talk with you about your cravings and try to help you to identify other things you might do instead of smoking.

What would be the best date and time to call for that session?

Document in Documentation Booklet

Could you also verify the phone number to call?

Document in Documentation Booklet

Thank you. Do you have any questions for me before we end our call? I look forward to speaking with you again soon.

## Rapport-Building

Begin by asking the participant how she and the baby are doing. Explain that this is the last PPCC call and that you have enjoyed speaking with her over the last few months.

#### **Documentation**

Go to the Documentation Booklet to complete initial questions. Based on responses, choose a topic to discuss from the list. This topic should be done last. If the participant has not quit smoking, you may wish to review her Quit Plan if she is willing to quit at this time or ask her which topic would be most helpful to review

For women who have not yet quit smoking:

Even though you haven't quit smoking completely, you have come a long way in learning more about yourself, why you smoke, and what steps you can take to fight the urge to smoke. The main focus of our last call is to offer you some additional tips on how to keep moving forward towards quitting smoking. Is there a topic that you would like to review to help you on your journey to quit smoking? If not, we can review your Quit Plan.

Coaches Notes: It is true that even after successfully quitting tobacco, there may be times that your client will be tempted to use tobacco products again. A certain situation or environment may trigger a craving weeks, months or even years after she has quit. The great news is that through this program, your client has learned the necessary techniques for conquering this addiction, and should she encounter challenges along the way, she can return to the behaviors and plans she used in this program to get back on track. Support your client by building her confidence in her successful quit and arming her with the knowledge that she can remain tobacco-free.

#### MAINTAINING A TOBACCO-FREE LIFE

Even if you have quit tobacco, there are still challenges that may arise. In this call, we will review some strategies to make sure you stay tobacco free.

Great job! You should now be well on your way to being tobacco-free. You have learned some terrific tips for staying quit and maybe even discovered a little more about yourself through your quit tobacco journey. The main focus from this point forward is to maintain your quit and continue your new, healthy lifestyle.

Here are some tips for continued success with maintaining your quit:

**Tip 1:** Practice constructive affirmations and be positive. If you find yourself dwelling on thoughts about using tobacco, you may be setting yourself up for a relapse. Change your thinking right away and remind yourself that you can stay tobacco-free. Reflect on the positive aspects of quitting and use the affirmations you learned at your 48-hour check in:

- "The craving for nicotine will pass whether I have some or not"
- "Having just one cigarette is not an option"
- "I am quitting one day at a time"
- "Using tobacco again is not an option"
- "I feel healthier when I don't use tobacco"
- "I will not let tobacco control my life"
- "I am an ex-tobacco user!"
- "I know quitting is difficult but the long-term benefits outweigh the short-term discomforts"
- "I am guitting for myself and for my new baby."

# List 3 new affirmations you are willing to try.

**Tip 2:** Always reward yourself for overcoming a trigger situation where in the past you would have used tobacco. Every time you make the choice not to use tobacco, you are reinforcing your commitment to yourself and a healthier life. The reward you use for these trigger situations can be as simple as allowing yourself an extra half hour to read a good book, a piece of chocolate, or something else you would truly enjoy.

## List 3 simple rewards you can use for overcoming trigger situations:

**Tip 3:** Add in some physical activity as a way to manage stress, anxiety, and improve your overall mood. It doesn't matter what you do, just move your body! Take a dance class, work in your garden, or start taking regular walks with a friend while pushing your baby in a stroller a few days a week for 30 minutes (even 15 minutes is great if you are just beginning or if it has been a while since you've been active). Once you get started, you can set goals to increase the time you spend doing your activity and add other types of movement that interest you. To help with this, you could wear a pedometer and count how many steps you're taking a day. The Healthy Mom, Healthy Baby program will provide you with one if you haven't received one already.

If you are already an active person, think of other activities that you can try and add them into your routine. Make your program well-rounded by including some resistance training and stretching. And finally, get full heart healthy benefits by increasing the duration of your physical activity to 60 minutes 4 to 6 days per week.

# Complete the following sentences to help you get started with or improve your level of physical activity:

I will do a scheduled activity on the following days (circle days you can commit to):

Monday Tuesday Wednesday Thursday Friday Saturday Sunday

I will be active for \_\_\_\_\_minutes each day

The best time of day for me to add in activity is:

Morning Lunch hour On work breaks After work After dinner

I will try this type(s) of physical activity:

My short-term physical activity goal is:

My long-term physical activity goal is:

**Tip 4:** Eat a healthy, well balanced diet. Be sure to review topic 9 regarding healthy eating. Include lots of fruits and vegetables that are in season, and even try a few new ones. Add adventure to your meals by trying new recipes, experimenting with herbs and spices, and taking the time to savor your creations.

Check out the following resources to help you get started with great cooking tips and delicious recipes:

www.foodnetwork.com www.eatingwell.com www.epicurious.com

**Tip 5:** Try a new hobby or class to dedicate your time to. This could be a class in which both you and your baby can participate. Since quitting tobacco, you may have noticed that you have extra time on your hands. Now is a great time to explore new areas of interest or to spend more time bonding with your baby. You can also do something positive for your community such as teach others to read through a local library program, volunteer at a neighborhood senior citizens' center, or start a walking group for new moms.

What are some new activities you are willing to try and how will you signup to participate?

**Tip 6:** Surround yourself with people who do not use tobacco. Use these people as a support system when you are having challenges, and ask them to join you in

one of your new activities. Think of the people in your life who you can spend time with and in what capacity.

Have confidence in the steps you have taken towards a healthier lifestyle. You now have the tools to remain an ex-smoker. Feel free to refer back to your quit plan during challenging times, or just as a refresher. You will need to remain vigilant in order to remain tobacco-free, but you can feel confident that you have taken the proper steps and that you are ready for any challenges that lie ahead. Congratulations on your great achievement!

**Tip to Quit:** Staying quit has nothing to do with luck or willpower. It is a matter of planning and commitment.

You have come a long way, and I want to congratulate you again on quitting smoking. It is a huge accomplishment, and I hope that this program has been helpful to you and can help you stay quit. Please remember that any time you have the urge to smoke or are craving a cigarette, you can call our toll-free number 24 hours a day 7 days a week through the end of 2014 and someone will be available to talk with you about your cravings and try to help you to identify other things you might do instead of smoking. After that, you can call 1-800-QUIT-NOW. Do you have any questions for me before we end our call? Thank you.

I can count on the following people to support me during my quit & I will let them know my plans by the following date:

<u>Name</u> <u>Date</u>

| I will also contact the following organizations or go to these websites by the following date: | |
|---|---|
| Organization/Website | <u>Date</u> |
| I plan to use the following support methods to hel | p me quit: |
| And, I have an appointment with my doctor on to determine which options best meet my needs. | |
| After careful consideration, I have decided the bes | st choice for me is to |
| ☐ Stop using tobacco all at once ☐ Gradually cut back the amount of tobacco by: cigarettes per day for the first week cigarettes per day for the second week cigarettes per day for the third week cigarettes per day for the fourth week | ζ. |

### **Countdown to Quit Week**

This section is designed to be completed every day, starting seven days out from your quit day. You will be given activities to do and tips to have a successful quit.

Coaches Notes: Now, it is action time. Your client is preparing her mind, her support team, and her environment for Quit Day. In the coming days and weeks, she will need additional support from you in order to feel prepared and confident for Quit Day. Encourage her to actively participate in all assignments and let her know that you are available for additional consultations if she has questions or concerns.

Today you are just 1 week away from freeing yourself from tobacco. Each day over the course of this next week you will check-in and complete individual daily assignments. In the previous weeks, the program has covered various tools and techniques to support you in your quit plan. Now we'll put what you've learned so far in action!

## **Day 7: Building Your Support**

Take this day to remind your support group that your quit date is nearing. Remember to include family, friends, co-workers, and neighbors. Call, email, write, meet in person...anything to let as many people as you can know that you are committed to quit!

| Assignment: List the people you will be telling today about your approaching quit date: | J |
|---|---|

### **Day 6: Exploring Positive Pleasures**

It's human nature to gravitate towards things we enjoy. If something feels good we are more likely to continue it, and if something feels bad we will probably stop. Quitting tobacco goes against your natural instinct to continue something that gives you pleasure. In order to successfully quit tobacco, it is important to find other things you enjoy to replace the positive feelings you get from tobacco.

| <b>Assignment:</b> Write down some alternative pleasures you can enjoy instrusing tobacco. Be sure to come up with some long- and short-term rewards a state of the st |
|---|
| meeting your goal to be tobacco-free. |

## Day 5: Plan Your Quit Day

You will likely feel some anxiety as your Quit Day approaches. It is a day you will look back on as the day that you became free from tobacco! Plan plenty of activities for this day so that you are occupied and distracted from the idea of using tobacco. Here are some suggestions to get you started Wash your car, carpets and drapes to clear them of the smell of tobacco smoke Go see a movie or go out for a meal in a smoke-free restaurant **Assignment:** Make a plan for your quit day full of healthy and productive activities that will distract you from using tobacco. Day 4: Show Me The Money! Lets face it, tobacco is using up your hard earned money every day. For most people, having some extra cash can be handy. Let's have a look at how much you will save when you're free of tobacco. packs/cans per day x 7 = (packs/cans per week) \_\_\_\_\_ packs/cans per week x \$\_\_\_\_(cost per pack/can)= \$\_\_\_\_(cost per week) \$ \_ (cost per week) x 52 = \$\_\_\_\_ (cost per year) You may also be aware that being a smoker can require you to pay more for medical insurance and life insurance. If you know how much more you are paying by being a smoker, make a note of it here: Medical insurance: additional\_\_\_\_\_ per month. Life insurance: additional per month. **Assignment:** What will you do with all the savings? List some things you can use the saved money on:

## Day 3: Creating a Tobacco Free Environment

The goal of this day is to remove ALL tobacco and related paraphernalia that will remind you of using tobacco once you quit. Gather these items in one area to be

tobacco cans, ashtrays, lighters, etc. The further away you are from tobacco and its accessories the more chance you'll have for success! Assignment: List the places where you keep tobacco related items that you will need to clean out: Check off the following items to throw away: Lighters and matches Ashtravs Tobacco company t-shirts, hats, and other items Clothing with cigarette burns Any loose cigarettes, extra packs of cigarettes or chewing tobacco **Day 2: Reviewing Your Motivation** It is common at this point to start to doubt that you will be able to guit or even that you want to guit. Refocus on the reasons why you are guitting tobacco and the benefits you will gain from doing so. Think about the health of your baby. Take a minute to write down your top three reasons for wanting to guit tobacco. **Assignment**: I am quitting tobacco for the following reasons: Day 1: 24 Hour Countdown Only 24 hours left! Tomorrow is the big day! Get out your quit plan and have it in an easily accessible place. Be sure to review everything on your plan once again to ensure that you are ready to take action. How are you feeling? Take a moment to jot down your feelings - both good and bad - about quitting tomorrow.

ready to throw away on quit day. Be sure you get all cigarettes, smokeless

| <b>Tip to Quit:</b> Try not to look at quitting as giving something up. Instead, look at al the positive things you will gain from quitting such as saving money, time, improving your health and your baby's health, and a tobacco-free life! |
|---|
| Assignment: Go through the following checklist to be sure that you have done everything you need to do to prepare for tomorrow: |
| <ul> <li>Reviewed your Personal Quit Plan</li> <li>Gathered ALL tobacco, ashtrays, lighters, etc. from your home, car, and work to throw away after your last cigarette today.</li> <li>Memorized your reasons for quitting tobacco that you listed in your quit plan</li> <li>Reminded at least two people that your quit day is tomorrow. Remember, the more support the better!</li> <li>If you will be using nicotine gum, patch, inhaler, or lozenge have them ready to use tomorrow morning.</li> <li>If you are going to attend any other support groups have a schedule of when and where they meet</li> <li>Be positive and have confidence that you CAN quit!</li> </ul> |

#### **Quit Week**

Today is the day you quit tobacco for good!

Your Quit Day: Congratulations!!! You made it to your quit day and are officially embarking on your journey to become tobacco-free! Be kind to yourself and make sure to do something special to mark the beginning of your new life. Here are some great things to try with space for you to add your own ideas:

- Perform a ceremony to mark the beginning of your journey
- Take your baby out for a special outing
- Buy a new DVD or CD with the money you save today
- Put it in writing fill out the quit tobacco contract at the end of this section to show your commitment to living a tobacco-free life
- Get a massage
- Start a journal

| • |
|---|
| _ |
| • |

Another great way to affirm the healthy lifestyle you are beginning is to recall the ways in which your body is already benefitting from being nicotine and smoke-free. You may remember these facts from our first call:

- 20 minutes after quitting, your blood pressure and heart rate drop
- 12 hours after quitting smoking your carbon monoxide levels drop to normal

As you travel further down the quit tobacco path, the physical benefits that you will reap become even more plentiful. Today is just the start!

Activate Your Quit Plan: Hopefully you are feeling excited about the quit plan you created; however it is perfectly normal to have some mixed emotions as well. To help bolster your confidence, keep a copy of your plan with you as a reminder of your goals. Now is the time to put all aspects of your plan into action. Call or see the people you listed as being supporters. Make sure you have removed all tobacco-related items from your house, office, and car. If you have decided to use an NRT, start using it today to help prevent cravings.

| Take some time to write down your thoughts and feelings day. What challenges do you think you might have today and overcome them? Is there anything you want to add to your qui | l how can you |
|---|---|

Create New Behaviors and Avoid Triggers: As you are aware from previous calls, one of the components of quitting tobacco is to create new behaviors that help break the association you have between tobacco and everyday routines. For example, if you always have a cigarette with your coffee, drink a different beverage like tea, or if you exit your workplace from the same door every time to go and smoke, choose a different exit and go for a walk instead.

In your quit plan, you created a list of triggers and thoughts that lead to the urge to use tobacco as well as a list of alternatives. In addition, you spent time identifying activities that contribute to smoking. **The focus for today is to stay busy and minimize your exposure to nicotine triggers!** Do anything to distract yourself, especially whenever a craving hits. Spend the day with your baby, go for a run or walk, drink a glass of water, suck on a mint, do 10 pushups, have a healthy snack, go see a movie, visit a friend, go shopping, or think about why you want to quit. Make sure to avoid situations that may trigger your urge to smoke such as bars or other places where other people are using tobacco.

| What are some changes to your routine that you will enact for at least the next few days? | |
|---|---|
| | _ |
| | _ |

At the End of Your Quit Day: Feel proud of your efforts and share the good news that you have been tobacco-free for 1 day!!! The first day is typically the hardest, but you did it! Although you may not feel mentally or emotionally at your best, your physical body is already repairing itself from the effects of nicotine and other by-products of long-term tobacco use. Here are some tips to help you end your day and set yourself up for success for the rest of the week:

- ✓ Have a nourishing meal that includes vegetables, healthy protein and a whole grain
- ✓ Spend time reviewing the reasons you are quitting and the benefits you will receive
- ✓ Relax by doing breathing exercises, stretches, or reading a good book
- ✓ Review your quit plan and prepare for tomorrow
- ✓ Be grateful for your body and your health

**48 Hours Tobacco Free:** Two days smoke free...what a great accomplishment! After about 48 hours of quitting tobacco your sense of smell and taste improves. Keep yourself motivated by taking notice of these changes. During the next day

be sure to smell something fragrant like flowers and eat a meal rich in spices to see if you notice the difference.

It is common at this point to feel a little overwhelmed and nervous. Maybe you are experiencing withdrawal symptoms due to the physical addiction to nicotine. It is normal to feel irritable, sad, nervous, and to have difficulty sleeping. These are indicators that your body is doing its job and clearing out the nicotine, and these sensations will pass. Stick with your quit plan...you will do great! Below is a list of things that you can do to increase your chances of success. Place a check next to the activities that you are currently doing:

| ☐ Drinking water | Asking for support |
|------------------------------------|-------------------------------|
| ☐ Using NRT/medication as directed | Reviewing my contract |
| ☐ Eating at regular intervals | Distracting myself from urges |
| ☐ Being physically active | Using my quit plan |
| ☐ Abstaining from alcohol | Managing stress |
| ☐ Noticing positive changes | Staying busy |
| ☐ Using website/program support | Positive self-talk |

In case you haven't been using positive self-talk up to this point, now is a good time to review some phrases that you can use for yourself:

- "The craving for nicotine will pass whether I have some or not"
- "Having just one cigarette is not an option"
- "I am quitting one day at a time"
- · "Using tobacco again is not an option"
- "I feel healthier when I don't use tobacco"
- "I will not let tobacco control my life"
- "I am an ex-tobacco user!"
- "I know quitting is difficult but the long-term benefits outweigh the short-term discomforts"

End today much like yesterday by taking some time to relax, review the strategies for success that you will use tomorrow, and get some quality sleep. Keep thinking about the reward you may have promised yourself once you have quit, and if that reward seems like a long way off, consider setting some short-term goals and rewards that reflect the smaller steps you are taking along the way.

One Week Tobacco Free: You did it! You are well on the road to staying tobacco-free. While it may not have been an easy week, you made it through. And, if you did have a slip and used tobacco, don't give up! Revise your plan and keep moving forward. This is a good time to reflect on the last 7 days and assess what worked and what adjustments you need to make to your plan for the weeks to come.
| How s | uccess | ful were | you exe | ecuting yo | ur quit | plan thi | s week? | | |
|---|---|---|---|---|---|---|---|---|---|
| 0% | ; | 20% | 409 | % | 60% | | 80% | | 100% |
| On a s | scale of | 1-10, ho | ow challe | enging did | you fir | nd the la | ıst week? | | |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| Not<br>challer | ot Challengi<br>nallenging | | | Challenging | 9 | | | | emely<br>enging |
| | | | | ner, what w<br>overcome | | biggest | challenge | s you fa | aced |
| | | | | ee over the | | 0 | 11 | | |
| them? | | | | | | | | | |
| On a s | scale of | <sup>-</sup> 1-10, ho | ow confi | dent are ye | ou that | you car | n stay qui | t? | |
| 1<br>Not<br>Confid | 2<br>ent | 3 | 4 | 5<br>Confident | 6 | 7 | 8 | | 10<br>remely<br>nfident |
| | | | | ow, what co<br>ress these | | | taying quit | do you | I<br> |

| How successful were you at starting new habits to take the place of using tobacco this week? | | | | | |
|---|---|---|---|---|---|
| 0% | 20% | 40% | 60% | 80% | 100% |
| with the mo | st (emotiona | ıl, triggers, cra | , what are the are<br>ivings, etc.), and<br>make new behav | what changes d | |
| Include how | v you feel ph | ysically and e | ou noticed about<br>motionally, imme<br>el good about! | | |
| give in to th | | he trick is to r | ays go away, reg<br>efocus your atter | | |
| takes about | t 3-4 days fo | r nicotine to le | common withdra<br>eave your system<br>check next to the | , so these withdr | awal ُ |
| Nervous Sadness Constan | ation<br>concentrati<br>ness<br>or depressi<br>t Cravings | | | | |
| | <b>-</b> | lings and acce | ept them, but kno | w that they will le | essen as |

# My Plan to Stay Tobacco-Free

| I officially became tobacco-free myself at regular intervals for on | on<br>ne vear to celebra | and will reward<br>te my ongoing success! |
|---|---|---|
| Time Tobacco-Free | Reward | io my engemig eneces. |
| 1 week | Newaru | |
| 1 month | | |
| 3 months | | |
| 6 months | | |
| 9 months | | |
| 1 year | | |
| I will also give myself the followi trigger situations: | ng small rewards | when I successfully overcome |
| I am making, or plan on making,<br>healthier lifestyle: | the following pos | sitive changes to support my |
| ☐ Being physically active at least | 30 minutes most d | ays of the week |
| ☐ Drinking 6-8 cups of water each | ı day | |
| ☐ Starting a new hobby or joining | a new group in my | community |
| ☐ Managing stress more effective | ly | |
| ☐ Eating well-rounded and nutrier | nt rich meals | |
| Reviewing my quit plan and cor | ntacting my suppor | t people if I feel tempted |
| ☐ Using healthy strategies to man | | |
| ☐ Doing some form of meditation | | |
| ☐ Eating breakfast most days of the | J | |
| My goal is to be physically active | e days p | er week for |
| minutes each time. The activitie | s/exercise(s) I wil | l do is/are |
| I will have decided to try the follo | | y,, on |
| the following date | | |

**Assignment:** What are your personal stressors and do you currently use tobacco products to cope with them? Examine the stress in your life this week and practice coping without the use of nicotine.

| Personal stressor | My typical reaction | What to try this week instead |
|-------------------|---------------------|-------------------------------|

# **APPROACHES TO QUITTING SMOKING**

This information is included in the Healthy Mom, Healthy Baby Guide and details various approaches to quitting smoking. You may reference this should the participant request additional information.

# Nicotine Replacement Therapy and Quit Smoking/Tobacco Prescriptions

You may have used a variety of methods if you have tried to quit tobacco in the past but to increase your chances of long-term success, you might be interested in exploring some additional support. There are numerous options for nicotine replacement therapies (NRTs) and prescription medications to help you quit. For many people, using these tools can substantially increase the chances of quitting tobacco. However, it is important to note that some of these may not be recommended for women who are pregnant or breastfeeding. It is essential that you discuss the use of any NRT or medication with your doctor.

✓ While developing your personal quit plan, you'll need to speak with your doctor and think ahead about which, if any, NRT or prescription you will use in order to have them available as your quit date approaches.

# **Nicotine Replacement Therapy (NRT):**

### **How Do NRTs Work?**

The function of an NRT is to replace the nicotine you get from cigarettes or smokeless tobacco products with nicotine from the NRT, but without the cancer-causing or toxic chemicals. Some NRT products are designed so that the amount of nicotine supplied is decreased in stages, thereby weaning the body of its dependence on nicotine and decreasing withdrawal symptoms. Nicotine withdrawal symptoms usually start within a few hours of quitting and can last for a few days to a few weeks. Symptoms of nicotine withdrawal include irritability, difficulty concentrating, feelings of depression, difficulty sleeping, increased appetite, cravings for nicotine, and headaches. NRTs help to relieve these symptoms by giving your body nicotine in amounts large enough to keep the symptoms at bay but small enough to help you break the nicotine craving cycle. By slowly tapering off nicotine, new behavioral skills can be learned to live a successful tobacco-free life.

### Types of NRT

NRTs are available over the counter in the form of a patch, gum, and lozenge. NRTs are also available by prescription from a doctor as an inhaler and nasal spray. **Always consult your doctor before taking any NRT.** 

| NRT | Description | Pros | Cons | Available over the counter |
|---|---|---|---|---|
| Nicotine Patch | A small band-aid like patch is worn on the body and releases a steady amount of nicotine that is absorbed through your skin and enters into the bloodstream. | Easy to use, private, available without a prescription, reduces nicotine withdrawal symptoms, doubles chances of quitting. | Somewhat costly. Can cause a rash at application site in some individuals. May cause vivid dreams. | Yes |
| Nicotine Gum | Nicotine gum supplies the body with nicotine to prevent sudden nicotine withdrawal symptoms. The nicotine released by the gum is absorbed through the lining of your mouth and into your bloodstream. | Good for people who find they need to do something with their mouth which makes it an excellent choice for smokeless tobacco users. Reduces nicotine withdrawal symptoms. Can be used to treat urges and cravings in an emergency and allows you to customize your nicotine level. Available in lots of flavors. | Must be chewed correctly and at regular intervals to fully benefit. Somewhat costly. | Yes |
| Nasal spray | Nicotine nasal spray comes in a pump bottle and is sprayed into the nose, one nostril at a time. Once the nicotine is on the nasal lining, it is absorbed into the bloodstream and delivered to the brain. | Quickly reduces nicotine cravings. Delivers nicotine faster than other products. | Cannot be used by allergy sufferers. Somewhat costly. May cause nose and throat irritation initially. It is possible to become dependent upon the spray. Some people may be uncomfortable using it in public. | No |
| Lozenges | Nicotine lozenges are slowly dissolved in the mouth to provide a dose of nicotine to your body via the lining of your mouth. There are two available strengths – 2mg and 4mg – depending on the amount of nicotine you currently take in. | Good for people who find they need to do something with their mouth which makes it an excellent choice for smokeless tobacco users. Reduces nicotine withdrawal symptoms. Available in two strengths to customize your nicotine dose. | Using too many lozenges in a short period of time can cause hiccups, heartburn and nausea. | Yes |

| Inhaler | The nicotine inhaler is placed in the mouth and administers the medication directly into the lung. The nicotine turns into vapor as it is inhaled, and is quickly absorbed into your bloodstream. | Easy to use. Wards off nicotine withdrawal symptoms and cravings by delivering nicotine quickly. | Somewhat costly. May cause mouth and throat irritation and a cough during first week of use. May cause stomach upset. | No |
|---|---|---|---|---|
| Varenicline<br>(Chantix) | Varenicline is the newest smoking medication and is available by prescription only. Varenicline targets nicotine receptors in the brain and blocks nicotine from attaching to the receptors, thereby reducing or eliminating the urge to use tobacco. Chantix is usually taken one to two weeks before your quit date and up to 11-12 weeks after quitting and helps in the quitting process. | Easy to use. Does not contain nicotine. Is not addictive. | Can have side effects such as nausea, sleep disturbance, constipation, gas, vomiting. Is costly and often not covered by insurance. Not recommended if breastfeeding. | No |
| Bupropion<br>(Wellbutrin,<br>Zyban) | Bupropion is a nicotine-free pill that acts on the brain by attaching to the same receptors that nicotine does to decrease urges. | Doubles chances of quitting, decreases your urge to smoke, is safe for most people, treats depression, can be used in combination with another NRT. | Somewhat costly, though a generic version is available and cheaper. May cause psychiatric side effects. | No |

# Which NRT Is Right For Me?

**Nicotine Patches:** A small band-aid like patch is worn on the body and releases a steady amount of nicotine that is absorbed through your skin. The nicotine enters into the bloodstream and is then delivered to specific places in the brain called receptors. The nicotine is released 24 hours a day in a smaller, less intense dose than you receive when smoking or using smokeless tobacco. Typically, nicotine patches are available in two dosages: 21 mg, which is recommended for people who smoke more than 10 cigarettes per day, or 14 mg, which is recommended for people who smoke less than 10 cigarettes per day. A final dose of 7mg is available for the final quit period. The dosage and the length of use of each dose are decreased according to the manufacturer's instructions or the plan you have created with your health care provider. Nicotine patches are generally available over the counter at your local pharmacy or for purchase over the internet.

**Pros:** Easy to use, private, available without a prescription, tames withdrawal symptoms, doubles chances of quitting, can be combined with other quit-smoking methods.

**Cons:** Somewhat costly. Can cause a rash at application site in some individuals. May cause vivid dreams.

**Nicotine Gum:** Nicotine gum supplies the body with nicotine to prevent sudden nicotine withdrawal symptoms and to allow you to wean off of nicotine. The nicotine released by the gum is absorbed through the lining of your mouth and into your bloodstream. This product is also available over the counter and comes in two dosages: 4mg, which is recommended for people who smoke 25 or more cigarettes per day, or 2 mg, which is recommended for people who smoke less than 25 cigarettes per day. The dosage and the frequency of use are decreased according to the manufacturer's instructions or the plan you have created with your health care provider. Nicotine gum is generally available over the counter at your local pharmacy or for purchase over the internet.

**Pros:** Good for people who find they need to do something with their mouths which makes it an excellent choice for smokeless tobacco users. Prevents nicotine withdrawal symptoms. Can be used to treat urges and cravings in an emergency and allows you to customize your nicotine level. Available over the counter and in a variety of flavors.

**Cons:** Must be chewed correctly and at regular intervals to fully benefit. Somewhat costly.

**Nicotine Lozenges**: Nicotine lozenges are slowly dissolved in the mouth to provide a dose of nicotine to your body. There are two available strengths – 2mg and 4mg – depending on the amount of nicotine you currently take in. This

medication is available over the counter and all dosing instructions on the package should be followed.

**Pros:** Easy to use. A good choice for smokeless tobacco users who are looking for an oral substitute.

**Cons:** Using too many lozenges in a short period of time can cause hiccups, heartburn and nausea.

**Nicotine Nasal Spray:** Nicotine nasal spray comes in a pump bottle and is sprayed into the nose, one nostril at a time. Once the nicotine is on the nasal lining, it is absorbed into the bloodstream and delivered to the brain. The nicotine effect is similar to smoking a cigarette or using a smoke-free tobacco product. Because of this immediate nicotine delivery, it is a good option for people who have a high dependence on nicotine. Guidelines for using this medication are provided by your health care provider. **This medication is available by prescription only.** 

**Pros:** Quickly reduces nicotine cravings. Delivers nicotine faster than other products.

**Cons:** May not be appropriate for allergy sufferers. Somewhat costly. Can be tricky to use properly. May cause nose and throat irritation for the first week. It is possible to become dependent upon the spray. Some people may be uncomfortable using it in public.

**Nicotine Inhaler:** The nicotine inhaler is placed in the mouth and administers the medication directly into the lung. The nicotine turns into vapor as it is inhaled into your lungs and is quickly absorbed into your bloodstream. **This medication is available by prescription only** and should only be used as directed by your health care provider.

**Pros:** Easy to use. Wards off nicotine withdrawal symptoms and cravings by delivering nicotine quickly.

**Cons:** Somewhat costly. May cause mouth and throat irritation and a cough during first week of use. May cause stomach upset. It is possible to become dependent on the dose of nicotine provided by the inhaler.

# Important Points Regarding the Use of NRT

NRT can be started as soon as you stop using tobacco. It should be used on a regular basis and according to the directions given by the manufacturer and your doctor. Starting and stopping the NRT will decrease the effectiveness of the therapy. For the best chance of quitting and staying quit, use NRT for at least 8-12 weeks. During the later weeks, the dosage of NRT is usually decreased until it

is completely stopped. This process allows the nicotine to be gradually tapered off so that the side effects of nicotine withdrawal will be lessened. **Be sure you have quit using tobacco before using an NRT to avoid a nicotine overdose**.

Always consult your doctor or health care provider before using any NRTs, especially if you are pregnant or breastfeeding, have heart disease, high blood pressure, stomach ulcers, or take insulin for diabetes.

# **Prescription Quit Smoking/Tobacco Medications:**

# **How Do Quit Smoking/Tobacco Medications Work?**

Prescription quit smoking/tobacco medications do not provide the body with nicotine as NRTs do. Instead, these medications target receptors in the brain to eliminate cravings. There are two primary types of medications which work differently in the body:

- The first type of medication helps to manage cravings by increasing the levels
  of certain feel good chemicals in the brain so that the urge for nicotine is
  decreased.
- The second type of medication targets the areas of the brain that nicotine goes
  to when it is delivered to the brain. The medication acts by sitting in these
  nicotine receptor sites, thus preventing nicotine from being able to enter and
  eliminating the usual nicotine rush that you get when smoking or using
  smokeless tobacco.

# Which Quit Smoking/Tobacco Medication is Right for Me?

Only your health care provider can determine which medication might be best for you as they may not be safe for individuals with certain health conditions. Planning ahead is crucial due to having to see your doctor first, and these medications generally need to be started a couple of weeks prior to your quit date in order to work optimally. As with the NRTs, quit smoking/tobacco medications are most effective when used in conjunction with a tobacco cessation plan and/or a structured support program.

# Types of Quit Smoking/Tobacco Medications

Tobacco cessation help is available through several prescription drugs. These medications are available in pill form only.

Varenicline (U.S. brand name - Chantix): Varenicline is the newest smoking medication and is available by prescription only. Varenicline targets nicotine receptors in the brain and blocks nicotine from attaching to the receptors, thereby reducing or eliminating the urge to use tobacco. Varenicline is usually taken one

to two weeks before your quit date and for up to 11-12 weeks after quitting. This medication cannot be used in combination with NRT. Varenicline is available by prescription only and should be used as recommended by your health care provider.

**Pros:** Easy to use. Does not contain nicotine. Is not addictive.

**Cons**: Can have side effects such as nausea, sleep disturbance, constipation, gas, vomiting. Is costly and often not covered by insurance. Is not recommended for women who are breastfeeding, and is only recommended during pregnancy when benefits outweigh risks (as determined by your doctor).

**Bupropion (U.S. brand names - Wellbutrin, Zyban):** Bupropion is a nicotine-free pill that acts on the receptor sites of two brain chemicals, norepinephrine and dopamine, allowing more of these chemicals to be present in the brain. Although the process by which this medication works is not entirely understood, research has repeatedly shown that people have a reduced desire to use tobacco while taking Bupropion. Planning ahead is important because you should start taking the medication before you stop using tobacco and continue taking it for about 12 weeks. Bupropion is available by prescription only and should be used as recommended by your health care provider.

**Pros:** Decreases your urge to smoke. Is safe for most people. Can be used in combination with NRT.

**Cons:** Somewhat costly, may cause side effects in some people such as anxiety, irritability, depression, suicidal thoughts, insomnia, constipation or dry mouth.

# <u>Important Points Regarding the Use of Prescription Quit Smoking/Tobacco</u> Medications

Quitting smoking/tobacco medications require a prescription from your doctor. It is important to take the medication only as prescribed. In order to be most effective, this medication should be started 1-2 weeks before your quit date. Make sure you see your doctor before your quit date and provide them with accurate health information so they can determine if taking a medication to quit is safe for you. Report any problems or troublesome side effects to your doctor as soon as they occur.

#### Alternatives to NRT and Medication

Nicotine replacement therapies are not for everyone, and there is some uncertainty about whether or not to use them during pregnancy or while breastfeeding. You may be interested in taking a different approach without nicotine or medications. Fortunately, there are various support groups, alternative therapies, and programs to help you in becoming tobacco-free. Many of the methods discussed below can be used in combination, and in conjunction with an NRT or prescription medication. Please note, however, that research has not shown these methods to be effective in smoking cessation.

# **Programs and Support Groups**

You might be able to find tobacco-free community programs or support groups in the Baltimore area. Whether it's through a hospital, community center or church, you'd be surprised at the resources around you. There are also plenty of groups and programs available online. In fact, certain websites are also a great way of finding groups in your neighborhood.

#### **Baltimore Resources**

- Freedom From Smoking® Class this free seven week program uses a positive behavior change approach, and helps participants develop their own plan on how to quit. In eight 90-minute sessions, you'll learn about reducing stress, cravings, and withdrawal symptoms, and how to control your weight while resisting the urge to smoke. To get information on when the next session starts, call 410-887-3828.
- Tobacco use Prevention and Cessation Program call 410-887-3828 to speak with a staff member. They offer free nicotine replacement gum, lozenges, smoking cessation classes and support.
- Baltimore City Health Department provides free smoking cessation group therapy and patch therapy
- **Good Samaritan Hospital** offers a smoking cessation support group that meets weekly, Mondays 6:30pm-8pm
- women.smokefree.gov

#### Meditation

If you are like most people, your tobacco use probably increases when you are under a lot of stress. It is important to find alternative ways to channel your stress when quitting tobacco and avoiding relapses. Meditation is one of the tools that can be used to help improve your ability to manage stress. There are many styles of meditation but the overall objective is the same...turn off your thoughts and experience deep relaxation. Once you develop a meditation practice, the benefits are long lasting and cumulative.

# **Putting it to ACTION:**

- For people new to this practice, you may want to be walked through the
  process with a guided meditation through a CD. There are also a variety of
  DVDs available. These products can be purchased at bookstores, at a variety
  of websites, or borrowed from your local library.
- Attend a class with an instructor to guide you through Yoga, Qi Gong or Tai
   Chi. If you can't find a class or if it is not feasible financially, you can purchase
   a DVD or borrow one from your local library and do it in the privacy of your
   own home.
- Deep breathing, imagery, progressive relaxation, walking meditation, prayer, and reading are all ways that you can meditate.

# **Aromatherapy**

Different smells can make you happy, sad, excited, irritated or relaxed. In aromatherapy, fragrant oils are used to calm and relax. Scents like lavender, cedar, eucalyptus, citrus, and tea tree are all commonly used for aromatherapy. Aromatherapy is often used in alternative medicine to reduce nausea, pain, and stress.

### **Putting it to ACTION:**

- Start and/or end your day with a warm bath. Add your fragrance of choice to the bath water and enjoy some time for yourself.
- You can find aromatic oils at health food stores and in a variety of shops that carry personal care items.
- Some aromatic oils such as peppermint can be applied directly to your wrist and temples to relieve stress.

# **Hypnosis**

Also referred to as hypnotherapy, hypnosis is a process whereby a trained hypnotherapist will guide you into a light trance. While in this state of mind, your practitioner will offer quit smoking suggestions that help to eliminate the urge to smoke. This therapy is also used to help people change negative behaviors and ease the symptoms of various health conditions.

Hypnotherapy works well for some individuals (especially those who struggle with willpower type thinking) and is not as effective for others. The length of treatment also varies, where some people receive benefit after one session while for others, it takes up to four sessions. For the best outcome, work with a hypnotherapist who specializes in tobacco cessation treatment.

### Acupuncture

Acupuncture is a Chinese medical treatment that was developed hundreds of years ago and has become increasingly popular around the world. During a session, the acupuncturist places thin needles into specific areas throughout the body called meridians. It is believed that the meridians are the channels where Qi or energy flows through the body. The objective of acupuncture is to improve the flow of energy in the body, which in turn restores balance and the body's ability to heal itself. Typically patients would visit the acupuncturist 1-2 times per week for up to 12 sessions or more.

**Tip to Quit:** While some of the methods in this session may be unfamiliar to you, it is important to keep an open mind. Being willing to try new things may provide you with just the support you need to succeed in your journey.

# **Progressive Relaxation Exercise**

Below is a script to follow to make this form of meditation a breeze. You can memorize the basic steps, create a voice recording that you can play during your designated meditation time, or do a guided progressive relaxation online (an example can be found here: <a href="http://www.youtube.com/watch?v=HFwCKKa--18">http://www.youtube.com/watch?v=HFwCKKa--18</a>)

Sit in a comfortable chair – reclining arm chairs are ideal. Lying on a bed is okay too. Get as comfortable as possible – no tight clothes or shoes and don't cross your legs. Take a deep breath; let it out slowly. You will be alternately tensing and relaxing specific groups of muscles. After tension, a muscle will be more relaxed than prior to the tensing. Concentrate on the feel of the muscles, specifically the contrast between tension and relaxation. In time, you will recognize tension in any specific muscle and be able to reduce that tension.

Don't tense muscles other than the specific group at each step. Don't hold your breath, grit your teeth, or squint. Breathe slowly and evenly and think only about the tension-relaxation contrast. Each tensing is for 10 seconds; each relaxing is for 10 or 15 seconds. Count "1,000 2,000..." until you have a feel for the time span. Note that each step is really two steps — one cycle of tension-relaxation for each set of opposing muscles.

Do the entire sequence below once a day until you feel you are able to control your muscle tensions. Be careful: If you have problems with pulled muscles, broken bones, or any medical contraindication for physical activities, consult your doctor first.

- 1. **Hands**. The fists are tensed; relaxed. The fingers are extended; relaxed.
- 2. **Biceps and triceps**. The biceps are tensed (make a muscle but shake your hands to make sure not tensing them into a fist); relaxed (drop your arm to the chair). The triceps are tensed (try to bend your arms the wrong way); relaxed (drop them).
- 3. **Shoulders**. Pull them back (careful with this one); relax them. Push the shoulders forward (hunch); relax.

- 4. **Neck (lateral)**. With the shoulders straight and relaxed, the head is turned slowly to the right, as far as you can; relax. Turn to the left; relax.
- 5. **Neck (forward)**. Dig your chin into your chest; relax. (Bringing the head back is not recommended you could break your neck)
- 6. **Mouth**. The mouth is opened as far as possible; relaxed. The lips are brought together or pursed as tightly as possible; relaxed.
- 7. **Tongue (extended and retracted)**. With mouth open, extend the tongue as far as possible; relax (let it sit in the bottom of your mouth). Bring it back in your throat as far as possible; relax.
- 8. **Tongue (roof and floor)**. Dig your tongue into the roof of your mouth; relax. Dig it into the bottom of your mouth; relax.
- 9. **Eyes**. Open them as wide as possible (furrow your brow); relax. Close your eyes tightly (squint); relax. Make sure you completely relax the eyes, forehead, and nose after each of the tensings.
- 10. **Breathing**. Take as deep a breath as possible and then take a little more; let it out and breathe normally for 15 seconds. Let all the breath in your lungs out and then a little more; inhale and breathe normally for 15 seconds.
- 11. **Back**. With shoulders resting on the back of the chair, push your body forward so that your back is arched; relax. Be very careful with this one, or don't do it at all.
- 12. **Butt**. Tense the butt tightly and raise pelvis slightly off chair; relax. Dig buttocks into chair; relax.
- 13. **Thighs**. Extend legs and raise them about 6in. off the floor or the foot rest but don't tense the stomach; relax. Dig your feet (heels) into the floor or foot rest; relax.
- 14. **Stomach**. Pull in the stomach as far as possible; relax completely. Push out the stomach or tense it as if you were preparing for a punch in the gut; relax.
- Calves and feet. Point the toes (without raising the legs); relax. Point the feet up as far as
  possible (beware of cramps if you get them or feel them coming on, shake them loose);
  relax.
- 16. **Toes**. With legs relaxed, dig your toes into the floor; relax. Bend the toes up as far as possible; relax<sup>7</sup>.

Now just relax for a while. As the days of practice progress, you may wish to skip the steps that do not appear to be a problem for you. After you've become an expert on your tension areas (after a few weeks), you can concern yourself only with those muscle groups. These exercises will not eliminate tension, but when it arises, you will know it immediately, and you will be able to "tense-relax" it away or even simply wish it away.

# HANDLING DIFFICULT QUESTIONS AND STATEMENTS

ADAPTED FROM PREGNANCY AND POSTPARTUM QUITLINE TOOLKIT (2007)

#### Overview

Pregnant women who smoke typically have complex emotions and conflicting feelings of "quitting for the baby." The following dialogue provides examples of messages that can be used during such times, and can help you gain confidence in routinely addressing tobacco use during pregnancy and postpartum.

\*\*Disclaimer: These examples are not meant to provide decision-making around using specific therapies. Individual Counselor judgment should guide each

#### SMOKERS HAVE NORMAL BABIES

"I have a lot of friends who smoked during pregnancy and have healthy babies." [Or, "I had two normal babies, and I smoked with them."]

Response:

clinical encounter.

"All pregnancies are different and it's hard to predict how any baby will be affected. However, we know that any smoking during pregnancy is a risk for the baby's health, so the best thing you can do for your health and the health of the baby is to stop."

#### **LOW BIRTH WEIGHT**

"Smoking can cause low birth weight, so I'll have an easier delivery." Response:

"It can be dangerous for the baby to be smaller, and there can be more complications. Smokers can also have premature babies, and there's less chance that the baby can go home with you from the hospital."

### **CUTTING DOWN**

"I used to smoke a pack a day. Isn't it better now that it's only half a pack? Isn't it OK to cut down?"

Response:

"You should feel good about smoking less, but the best thing for your health and your baby's health is no cigarettes at all. Every cigarette gives your baby carbon monoxide. There is no safe cigarette. There are more and better ways these days to help people to stop smoking. We'd be happy to help you give it a try."

### **WEIGHT GAIN**

"I'll gain weight if I quit, and that's bad for the baby, right?"

"It sounds like weight is an important issue for you. Some smokers gain weight when they quit, but there are ways to make sure it's temporary. You should focus on getting healthy, and quitting can really help you do

that. Gaining weight during pregnancy and carrying extra weight after giving birth is normal, and is less harmful than continuing to smoke."

#### STRESS

"I am so stressed with having this baby, and smoking helps me relax. Won't the stress just get worse if I quit?"

Response:

"Smoking makes you think you're more relaxed, but cigarettes actually increase your heart rate and blood pressure. Can you think of other ways to relax that you might try instead? (taking a walk, a bath, calling a friend)

### **IRRITABLE**

"I get so irritable and crazy if I don't have a cigarette."

Response:

"It's completely normal to feel that way – it's your body's reaction to not having the nicotine. It's called nicotine withdrawal, and these symptoms will decrease over time. The important thing is to make a plan, and figure out what you can do instead of smoke. Tell me about the last time you stopped smoking . . ."

### **CRAVINGS**

"I get terrible cravings for cigarettes, like when my boyfriend is smoking." Response:

"These cravings are completely normal, and are a part of the dependence that happens with nicotine. It's like a hunger pain, though, and it can go away in a few minutes. It's important to distract yourself, and change your routine. What could you do differently when your boyfriend comes over and wants to smoke?"

# **PASSIVE SMOKE**

"My mom and boyfriend smoke around me. Isn't that bad for the baby?" Response:

"Yes, secondhand smoke is harmful to pregnant women as well as to infants and children. It sounds like you're thinking seriously about tobacco and smoking, which is great. What are your thoughts about asking them to not smoke at all inside the house or car?"

# FRIENDS SMOKE

"All my friends smoke. What am I going to do, stop seeing them?" Response:

"It sounds like it's hard for you when your smoking friends are around. It's OK to ask your friends not to smoke around you, for you and the baby. Most smokers don't mind if they're asked nicely to smoke somewhere else. It might also be a good idea to go to places where you can't smoke, like stores or certain restaurants."

#### AFTER PREGNANCY

"It wasn't too bad to quit while I was pregnant. Smoking made me a little nauseous. But I am smoking, now that I had the baby."

# Response:

"You quit smoking during your pregnancy, and you should be very proud of yourself. It can be hard to stop smoking, but you did it. Now that you're a mom, you have new responsibilities. But it's really important that you not smoke, for you as well as for your baby because it's bad for the baby's health to be around secondhand smoke too. Are you interested in trying to stop smoking again?"

### **USING MEDICATIONS**

"Last year I quit for a while with the patch. Can't I use that now?" (wants to quit) Response:

"Nicotine patches and gum can be very helpful with quitting smoking. But because you're pregnant/breastfeeding, you'll need to talk with your doctor about using them now. We can talk about some alternative approaches.

### **MULTIPLE RISK FACTORS**

"You're asking me to do so many things at once – eat better, exercise, stop smoking."

# Response:

"Actually, you're right. It is hard to make changes at the same time. What's important is that you plan for a change that's realistic and practical. Do you think that you could seriously try to stop smoking in the next 2 weeks?"

### **NEVER TOO LATE**

"It's really too late for me to quit now."

### Response:

"Your baby can benefit from quitting anytime, and it's still important to think about quitting. And there are many benefits of being a smoke-free mom. You'll be a better role model for your baby. Your own health will improve as well."

# **DEPRESSED**

"I'm afraid that when I quit smoking, like I did before, I'll feel down and depressed."

### Response:

"Nicotine can have powerful effects on your brain, including your mood. This can be a normal reaction to not having nicotine. It's important that we talk about this, and make sure we know how you're feeling after you stop smoking. It would also be a good idea to get some referrals from the social worker at the Maryland Women's Center."

# DISTRESSED PARTICIPANT PROTOCOL

If the participant displays distress during the call, you will administer the following distress protocol and then immediately contact a supervisor to report the situation. Keep in mind that respondent distress during the interview is different from respondent anger or frustration during the introduction and consent process. By "distress" we are referring to respondents who are most likely upset by the content of the session as it relates to their own personal experiences, versus an angry household member who is refusing to complete the call. The respondent distress protocol includes steps to follow for different levels of distress: mild, moderate, or severe distress.

# Step 1: Recognize that a respondent is possibly distressed.

The following are signs that may indicate a respondent is possibly distressed:

- Hesitancy to answer a question or questions;
- Refusal to answer questions or to continue the call;
- Lowering of the volume or tone of voice;
- Responding in an agitated manner by raising her voice or using inappropriate language;
- Crying;
- Indications of tremors, a quivering in the respondent's voice;
- Hearing the respondent tap her fingers, or an instrument on the telephone or surface; or
- Disorganization, dissociation, or non-responsiveness to questions asked.

# Step 2: Observe the level of distress that a respondent is apparently experiencing.

Below is a table that provides some guidance to an interviewer as to what indicators you might come across on the telephone indicating that a person may be in distress.

NOTE: The indicators listed below are examples - not an exhaustive list.

| LEVEL OF DISTRESS<br>MILD | SIGNS OR INDICATORS OF POSSIBLE DISTRESS • Change in voice tone or volume. • Hesitancy to answer questions. • Use of inappropriate language/cursing. • Provides non-relevant answers to questions asked. • Displays an unwillingness or hesitancy to continue. |
|---|---|
| MODERATE | MILD signs plus any of the following: • Displays signs of distress that may include long pauses, or sighing. • Sobbing, weeping, and/or crying on the telephone. • Displays flat voice tones. • Being non-responsive. • Provides nonsensical/bizarre answers. |
| SEVERE | • Talks about passive or active suicidal thoughts with or without a plan. • Talks about wishing another person was dead with or without a plan to kill the person. • Respondent asks for immediate help from emergency services or 911. • Respondent poses an immediate threat to themselves or someone else. |

# Step 3: Respond appropriately to the situation.

Based on your observation of the level of distress, it is imperative that you react appropriately and with sensitivity. When a respondent displays emotional distress, either verbally or non-verbally (i.e., crying) you should acknowledge their distress and if appropriate offer to finish the call at another time. Some acknowledgement phrases you may use include:

# **Acknowledgement Phrases**

- —It sounds like these questions may be upsetting to you. Would you like to take a short break and get a drink of water?
- —Would you like me to skip this question and go to the next section?
- —Are you ok? Do you want to keep going with the call? If not, I can call you back another time to finish.
- —Thank you for sharing that.
- —I know it must be difficult to talk about that.
- —I can tell that you're frustrated. Would you like me to call back at a better time to complete the interview?
- —Would you like to take a break and continue this at a later time?
- —I really appreciate you telling me this.

If the participant chooses to terminate the call because of distress, you should record detailed comments about the case as well as complete a problem sheet describing the distress, and then pass this information to your supervisor so that it can be reviewed by project staff. All such cases will be reviewed.

Similarly, in the unlikely event that a respondent exhibits severe distress by expressing thoughts/intentions of suicide, the interviewer will stop the interview and will encourage the respondent to call the National Lifeline (1-800-273-8255 (TALK)). You may also ask permission to call Lifeline with them on the line, then transfer them to that hotline. Detailed comments about any case involving suicide should be recorded in a problem sheet and immediately reported to your Supervisor and the Principal Investigator.